CLINICAL TRIAL: NCT02215096
Title: A Phase I, Open-label, Dose-finding Study of GSK2636771 Administered in Combination With Enzalutamide (Xtandi^TM ) in Male Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: Dose-finding Study of GSK2636771 When Administered in Combination With Enzalutamide in Male Subjects With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200331; 2013-005111-27 (EudraCT Number)
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Neoplasms
Keywords: enzalutamide; metastatic castration-resistant prostate cancer; GSK2636771; PI3K-beta; PTEN deficiency
MeSH Terms: conditions — Neoplasms | interventions — GSK2636771; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1-Dose Escalation (Experimental): Subject receiving a stable dose of enzalutamide 160 mg once daily will receive GSK2636771 following a modified 3+3 dose escalation procedure (Cohort -1: 200 mg, Cohort 1: 300 mg and Cohort 2: 400 mg) to evaluate the safety and PK for each combination dose level and to guide selection of the RP2D of the combination. If the combination doses in Cohort 1 are not tolerable, lower doses as defined in the de-escalation cohort (Cohort -1) will be evaluated. If the de-escalation cohort (Cohort -1) is not tolerable, further dose-escalation using a continuous daily dosing schedule for both compounds simultaneously will be terminated. Additional dose levels of GSK2636771 or alternative dosing schedules may be explored based upon ongoing assessment of safety and PK. Dose modification decisions will be made utilizing all available data at the end of each DLT determination period (28 days).
  Interventions: Drug: GSK2636771; Drug: Enzalutamide
- Phase 2- Dose Expansion (Experimental): Additional 20 subjects will be assigned to receive GSK2636771 at the MTD or RP2D determined in the Dose-Escalation Phase while continuing treatment with enzalutamide to evaluate the long-term safety of the combination as well as the 12-week non-PD rate
  Interventions: Drug: GSK2636771; Drug: Enzalutamide

INTERVENTIONS:
Drug: GSK2636771 — GSK is available as 100 mg hard gelatin oral capsule to be taken once daily/continuous until treatment withdrawal under fasting conditions for at least 1hour (h) before and 2h after dosing with approximately 200 mL of water
Drug: Enzalutamide — Enzalutamide will be sourced locally from commercial stock for sites in countries where it is approved

SUMMARY:
This Phase I, open-label, dose-finding, multicenter study is designed to determine the recommended Phase II dose (RP2D) for the combination of an orally administered Phosphatidylinositol-4,5-bisphosphate 3-kinase beta (PI3K-beta) inhibitor (GSK2636771) with enzalutamide. Subjects with phosphatase and tensin homolog (PTEN)-deficient metastatic castration-resistant prostate cancer (mCRPC) who are receiving a stable dose of enzalutamide with a recently demonstrated progression (either by RECIST [Response Evaluation Criteria In Solid Tumors] version 1.1, prostate-specific antigen [PSA] progression, and/or progression in bone) per the Prostate Cancer Working Group 2 (PCWG2) criteria will be enrolled. Eligible subjects will be enrolled in the Dose-Escalation Phase to determine the maximum tolerated dose (MTD) of the combination therapy using a modified 3+3 dose escalation procedure. The safety, pharmacokinetics (PK) and clinical efficacy will also be assessed to guide the selection of the RP2D. The starting dose will be GSK2636771 300 mg once daily in combination with the recommended dose (160 milligram [mg] once daily) of oral enzalutamide. Once the RP2D has been established, additional subjects will be enrolled in the Dose Expansion Phase to further evaluate the safety, PK and preliminary clinical activity. Safety assessments will be performed throughout the study including physical examinations, vital signs, clinical laboratory tests, 12 lead electrocardiograms and monitoring of adverse events. Blood samples will be collected for pharmacokinetic analysis. Subjects will continue treatment until an unacceptable toxicity, disease progression, withdrawal of consent or death occurs. A post-treatment follow-up visit will be performed within 30 days of the last dose of study treatment. Xtandi is a registered trademark of Astellas Pharma Inc

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent provided
* Males >=18 years of age (at the time consent is obtained)
* Histologically or cytologically confirmed diagnosis of prostate adenocarcinoma, surgically castrated or continuous medical castration (for >=8 weeks prior to Screening)
* Serum testosterone <50 nanogram per deciliter (ng/dL) (1.7 nanomole per liter [nM/L])
* PTEN deficient tumor as documented from archival or fresh (from biopsy) tumor tissue analyzed by GlaxoSmithKline selected laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Completed at least 12 weeks of prior continuous therapy with enzalutamide. A 2 week or less treatment (enzalutamide) holiday will be permitted prior to initiating study treatment.
* Most recent enzalutamide dose received is 160 mg once daily with no change in dose for at least 2 weeks prior to Screening.
* Has progressive disease at time of enrollment defined as one or more of the following criteria: PSA progression defined by PCWG2 criteria or soft tissue disease progression defined by RECIST 1.1 or bone disease progression defined by PCWG2 criteria Able to swallow and retain orally administered medication.
* Adequate baseline organ function.
* Must have a QT interval corrected for heart rate according to Fridericia's formula (QTcF) <470 milli seconds (msec) or <480 msec with bundle branch block.
* Male subject with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from time of Screening until 3 months after the last dose of study treatment.

Exclusion Criteria:

* Prior treatment with: anti-cancer therapy (e.g., chemotherapy with delayed toxicity, immunotherapy, biologic therapy or chemoradiation) within 21 days (or within 42 days if prior nitrosourea or mitomycin C containing therapy) prior to enrollment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to enrolment. Subjects may remain on luteinizing hormone releasing hormone (LHRH) agonists (i.e., leuprolide, goserelin, triptorelin or histrelin). Subjects must have prior enzalutamide treatment; Any PI3K, AKT or mammalian target of rapamycin (mTOR) inhibitors; Investigational drug(s) within 30 days or 5 half-lives, whichever is longer, prior to enrollment
* Prior malignancy other than CRPC. Subjects who have been disease-free for 5 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Current use of or anticipated requirement during the study of prohibited medication(s) (any investigational drug(s), Other anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy, or hormone therapy other than for replacement), AR antagonists (e.g., bicalutamide, flutamide, nilutamide), 5-alpha reductase inhibitors (e.g., finasteride, dutasteride), Androgens (e.g., testosterone, dihydroepiandrosterone), Herbal medication(s) that may affect PSA levels (e.g., saw palmetto), Other herbal medications including, but not limited to: St. John's wort, kava, ephedra (ma huang), gingko biloba, yohimbe and ginseng)
* Any unresolved >=Grade 2 (per CTCAE v 4.0) toxicity from previous anti-cancer therapy at the time of enrollment, except alopecia or Grade 2 anemia (if hemoglobin is >9.0 g/dL)
* Any >=Grade 2 hypophosphatemia (per CTCAE v4.0) at the time of enrolment
* Serum calcium >=Grade 1 (per CTCAE v4.0) at time of enrolment, unless ionized calcium is within normal range
* Presence of any clinically significant gastrointestinal (GI) abnormality or other condition(s) that may alter absorption such as malabsorption syndrome or major resection of the stomach or substantial portion of the small intestine
* Active peptic ulcer disease or history of abdominal fistula, GI perforation, or intra abdominal abscess within 28 days prior to enrolment
* Previous major surgery within 28 days prior to enrolment
* Known active infection requiring intravenous (IV) or oral anti-infective treatment
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screening (testing at time of screening is not required).
* A positive test for human immunodeficiency virus (HIV) antibody (testing at time of screening is not required).
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease)
* History of seizure or any condition that may predispose subject to seizure (e.g., prior cortical stroke or significant brain trauma). History of loss of consciousness or transient ischemic attack within 12 months of randomization
* History or evidence of cardiovascular risk including any of the following: Clinically significant electrocardiogram abnormalities including second degree (Type II) or third degree atrioventricular block; history of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, stenting, or bypass grafting within the past 6 months prior to enrolment, Class III or IV heart failure as defined by the New York Heart Association functional classification system, LVEF below 50%; known cardiac metastases
* Poorly controlled hypertension (defined as systolic blood pressure of>=150 millimeter of mercury (mmHg) or diastolic blood pressure of >100 mmHg based on a mean of three measurements at approximately 2-minute intervals)
* History of congenital platelet function defect (e.g., Bernard-Soulier syndrome, Chediak-Higashi syndrome, Glanzmann thrombasthenia, storage pool defect)
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2636771or enzalutamide or excipients.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dose of study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (6):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Houston, Texas
- United Kingdom (2):
  - GSK Investigational Site, London
  - GSK Investigational Site, Sutton

REFERENCES:
- [Derived] Sarker D, Dawson NA, Aparicio AM, Dorff TB, Pantuck AJ, Vaishampayan UN, Henson L, Vasist L, Roy-Ghanta S, Gorczyca M, York W, Ganji G, Tolson J, de Bono JS. A Phase I, Open-Label, Dose-Finding Study of GSK2636771, a PI3Kbeta Inhibitor, Administered with Enzalutamide in Patients with Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2021 Oct 1;27(19):5248-5257. doi: 10.1158/1078-0432.CCR-21-1115. PMID 34281912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, dose finding study of GSK2636771 administered in combination with Enzalutamide in male participants with Metastatic Castration-Resistant Prostate Cancer (mC-RPC) conducted at 7 centers across United Kingdom and United States.
Pre-assignment Details: A total 37 participants were enrolled in this study and entered in the enzalutamide run-in period, of which 36 participants received GSK2636771+enzalutamide and completed the combination treatment period (TP).
Groups:
- Enzalutamide Only (run-in Period): Participants received enzalutamide monotherapy at the approved dose of 160 milligrams (mg) once daily orally for 14 days in run-in period to achieve near-steady-state levels of enzalutamide prior to initiating combination therapy with GSK2636771. Participants who completed the enzalutamide run-in period continued with the combination therapy with GSK2636771.
- GSK2636771 200mg/Enzalutamide 160mg Escalation: Participants received GSK2636771 200 mg once daily orally in combination with enzalutamide 160 mg orally once daily in dose escalation cohort.
- GSK2636771 200mg/Enzalutamide 160mg Expansion: Participants received GSK2636771 200 mg once daily orally in combination with enzalutamide 160 mg orally once daily in dose expansion cohort. Participants were enrolled in this cohort as an expansion of the dose escalation cohort (GSK2636771 200 mg/ enzalutamide 160 mg) to collect adequate data on safety, pharmacokinetics and pharmacodynamics.
- GSK2636771 300mg/Enzalutamide 160mg Escalation: Participants received GSK2636771 300 mg once daily orally in combination with enzalutamide 160 mg orally once daily in dose escalation cohort.
- GSK2636771 400mg/Enzalutamide 160mg Escalation: Participants received GSK2636771 400 mg once daily orally in combination with enzalutamide 160 mg orally once daily in dose escalation cohort.
Period: Run-In Period (Up to Week 2)
Arm/Group | Enzalutamide Only (run-in Period) | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Started | 37 | 0 | 0 | 0 | 0
Completed | 36 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Period: Combination TP (Up to Maximum 654 Days)
Arm/Group | Enzalutamide Only (run-in Period) | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Started | 0 | 11 | 11 | 12 | 2
Completed | 0 | 9 | 10 | 10 | 1
Not Completed | 0 | 2 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Safety Population consisted of all participants who received at least one dose of GSK2636771 or Enzalutamide.
Groups:
- All Participants: Participant received enzalutamide monotherapy at the approved dose of 160 mg once daily orally for 14 days in run-in period to achieve near-steady-state levels of enzalutamide prior to initiating combination therapy with GSK2636771. In combination treatment period, participants received GSK2636771 200 mg or 300 mg or 400 mg once daily orally in combination with enzalutamide 160 mg once daily orally in dose escalation/ expansion cohorts.
Arm/Group | All Participants
Number analyzed (Participants) | 37
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0
  18-64 years | 9
  65-74 years | 20
  >=75 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1
  Asian-South East Asian Heritage | 1
  White-White/Caucasian/European Heritage | 34
  Native Hawaiian or Other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs) During run-in Period
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, protocol-specific SAEs: All events of possible study treatment-induced liver injury with hyperbilirubinemia defined as alanine aminotransferase (ALT) >=3 times upper limit of normal (ULN), and bilirubin >=2 times ULN (>35 percent [%] direct) (or ALT >=3 times ULN and international normalized ratio (INR) >1.5 if INR is measured) or termed 'Hy's Law' events (INR measurement is not required and the threshold value stated did not apply to participants receiving anticoagulants) or any new primary cancer.
Time Frame: Up to Week 2
Population: All Treated Safety Population consisted of all participants who received at least one dose of Enzalutamide.
Measure: Count of Participants; unit: Participants
Groups:
- Enzalutamide Only (run-in Period): Participants received enzalutamide monotherapy at the approved dose of 160 mg once daily orally for 14 days in run-in period to achieve near-steady-state levels of enzalutamide prior to initiating combination therapy with GSK2636771. Participants who completed the enzalutamide run-in period continued with the combination therapy with GSK2636771.
Arm/Group | Enzalutamide Only (run-in Period)
Number analyzed (Participants) | 37
Participants
  Non-SAEs | 11
  SAEs | 1

2. Primary Outcome: Number of Participants With Non-SAEs and SAEs During Combination Treatment Period
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participants, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, protocol-specific SAEs: All events of possible study treatment-induced liver injury with hyperbilirubinemia defined as ALT >=3 times ULN, and bilirubin >=2 times ULN (>35% direct) (or ALT >=3 times ULN and INR >1.5 if INR is measured) or termed 'Hy's Law' events (INR measurement is not required and the threshold value stated did not apply to participants receiving anticoagulants) or any new primary cancer.
Time Frame: Up to maximum 675 days
Population: All Treated Safety Population consisted of all participants who received at least one dose of GSK2636771 or Enzalutamide. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Participants
  Non-SAEs | 11 | 11 | 12 | 2
  SAEs | 2 | 2 | 2 | 0

3. Primary Outcome: Number of Participant With Dose-limiting Toxicities (DLT) During Combination Treatment Period
Description: An event was considered as DLT if the event was attributed (definitely, probably or possibly) to study treatment, occured within the first 28 days of combination treatment (DLT reporting period), and met one of the following criteria: Febrile neutropenia of any grade or duration as per Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, Grade 4 neutropenia lasting >5 days, Grade 3 or greater non-hematologic toxicity that cannot be controlled with routine supportive measures, Grade 4 thrombocytopenia, ALT >3 times ULN with bilirubin >2 times ULN or ALT >=3 times ULN and >=1.5 times Baseline ALT value, if enrolled with liver metastases/tumor infiltration at Baseline), together with bilirubin >=2 times ULN.
Time Frame: Up to Day 28
Population: All Treated Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Participants | 1 | 0 | 2 | 2

4. Primary Outcome: Percent Change From Baseline in Hematology Parameters During Combination Treatment Period: Basophils, Eosinophils, Hematocrit, Hemoglobin, Lymphocytes, MCH, MCV, Monocytes, Total Neutrophils, Platelet Count, WBC Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, hematocrit, hemoglobin, lymphocytes, mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), monocytes, total neutrophils, platelet count and white blood cells (WBCs) count. Baseline value is the latest GSK2636771 pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100 multiplied by (post-Baseline visit value minus Baseline divided by Baseline).
Time Frame: Baseline (Day 1), Weeks 2,3,4,5,8,12,16,20,24,28,32,36,40,44,48,52,56,60,64,68,72,76,80,84 and 88
Population: All Treated Safety Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Percent change
  Basophils, Week 2, n=5,4,5,1: number analyzed (Participants) | 5 | 4 | 5 | 1
  Basophils, Week 2, n=5,4,5,1 | 20.000 (103.6822) | 0.000 (0.0000) | 30.000 (48.0885) | 33.330 (NA) — Standard deviation could not be calculated for single participant.
  Basophils, Week 3, n=5,5,6,1: number analyzed (Participants) | 5 | 5 | 6 | 1
  Basophils, Week 3, n=5,5,6,1 | 0.000 (70.7107) | 27.500 (43.6606) | -16.270 (38.4859) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Basophils, Week 4, n=5,4,5,1: number analyzed (Participants) | 5 | 4 | 5 | 1
  Basophils, Week 4, n=5,4,5,1 | -16.666 (79.9314) | 25.000 (50.0000) | 26.666 (43.4612) | 33.330 (NA) — Standard deviation could not be calculated for single participant.
  Basophils, Week 5, n=4,4,5,0: number analyzed (Participants) | 4 | 4 | 5 | 0
  Basophils, Week 5, n=4,4,5,0 | -37.500 (94.6485) | 25.000 (50.0000) | 27.380 (46.9143) |
  Basophils, Week 8, n=4,4,4,0: number analyzed (Participants) | 4 | 4 | 4 | 0
  Basophils, Week 8, n=4,4,4,0 | -12.500 (25.0000) | 25.000 (50.0000) | 139.583 (188.2399) |
  Basophils, Week 12, n=3,4,3,0: number analyzed (Participants) | 3 | 4 | 3 | 0
  Basophils, Week 12, n=3,4,3,0 | 0.000 (100.0000) | 25.000 (50.0000) | 51.190 (42.3084) |
  Basophils, Week 16, n=3,4,1,0: number analyzed (Participants) | 3 | 4 | 1 | 0
  Basophils, Week 16, n=3,4,1,0 | -33.333 (57.7350) | 16.668 (33.3350) | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Basophils, Week 20, n=2,3,1,0: number analyzed (Participants) | 2 | 3 | 1 | 0
  Basophils, Week 20, n=2,3,1,0 | -50.000 (70.7107) | 0.000 (0.0000) | 50.000 (NA) — Standard deviation could not be calculated for single participant. |
  Basophils, Week 24, n=2,1,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0
  Basophils, Week 24, n=2,1,0,0 | -50.000 (70.7107) | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Basophils, Week 28, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Basophils, Week 28, n=1,0,0,0 | 100.000 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Basophils, Week 32, n=2,1,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0
  Basophils, Week 32, n=2,1,0,0 | 0.000 (141.4214) | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Basophils, Week 36, n=2,1,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0
  Basophils, Week 36, n=2,1,0,0 | -50.000 (70.7107) | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Basophils, Week 40, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Basophils, Week 40, n=0,1,0,0 |  | 100.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Basophils, Week 44, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Basophils, Week 44, n=0,1,0,0 |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Basophils, Week 48, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 52, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 56, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 60, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 64, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 68, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 72, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 76, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 80, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 84, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Basophils, Week 88, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Eosinophils, Week 2, n=9,8,8,2: number analyzed (Participants) | 9 | 8 | 8 | 2
  Eosinophils, Week 2, n=9,8,8,2 | -26.321 (47.4470) | -8.754 (30.6984) | -19.135 (47.3780) | -2.175 (3.0759)
  Eosinophils, Week 3, n=8,8,9,2: number analyzed (Participants) | 8 | 8 | 9 | 2
  Eosinophils, Week 3, n=8,8,9,2 | 13.085 (40.8232) | 13.994 (65.2691) | 4.704 (68.1450) | 54.350 (64.5588)
  Eosinophils, Week 4, n=8,8,8,2: number analyzed (Participants) | 8 | 8 | 8 | 2
  Eosinophils, Week 4, n=8,8,8,2 | 11.136 (36.6046) | -3.626 (75.4907) | 13.333 (57.7624) | -2.175 (3.0759)
  Eosinophils, Week 5, n= 7,7,8,1: number analyzed (Participants) | 7 | 7 | 8 | 1
  Eosinophils, Week 5, n= 7,7,8,1 | 54.970 (110.7083) | -23.809 (43.1487) | 9.708 (42.6803) | 100.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 8, n=6,7,8,1: number analyzed (Participants) | 6 | 7 | 8 | 1
  Eosinophils, Week 8, n=6,7,8,1 | 16.857 (53.6217) | 5.953 (32.8832) | 90.104 (102.6830) | -100.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 12, n=4,6,6,1: number analyzed (Participants) | 4 | 6 | 6 | 1
  Eosinophils, Week 12, n=4,6,6,1 | 31.250 (47.3242) | 1.390 (41.6394) | 72.578 (129.4696) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 16, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Eosinophils, Week 16, n=5,5,3,1 | 2.120 (15.8040) | -17.626 (34.2120) | 62.500 (119.2424) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 20, n=3,5,3,1: number analyzed (Participants) | 3 | 5 | 3 | 1
  Eosinophils, Week 20, n=3,5,3,1 | 9.090 (15.7443) | 15.000 (81.7340) | 66.667 (115.4701) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 24, n=3,3,2,1: number analyzed (Participants) | 3 | 3 | 2 | 1
  Eosinophils, Week 24, n=3,3,2,1 | 18.183 (31.4945) | -50.000 (66.1438) | 50.000 (70.7107) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 28, n=3,2,2,1: number analyzed (Participants) | 3 | 2 | 2 | 1
  Eosinophils, Week 28, n=3,2,2,1 | 44.950 (63.9644) | -87.500 (17.6777) | 0.000 (141.4214) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 32, n=4,2,2,1: number analyzed (Participants) | 4 | 2 | 2 | 1
  Eosinophils, Week 32, n=4,2,2,1 | 589.773 (1140.3590) | -25.000 (106.0660) | 0.000 (141.4214) | -100.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 36, n=3,1,2,1: number analyzed (Participants) | 3 | 1 | 2 | 1
  Eosinophils, Week 36, n=3,1,2,1 | 13.890 (24.0582) | 50.000 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (141.4214) | 100.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 40, n=1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Eosinophils, Week 40, n=1,1,1,1 | 100.000 (NA) — Standard deviation could not be calculated for single participant. | 125.000 (NA) — Standard deviation could not be calculated for single participant. | 100.000 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Eosinophils, Week 44, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Eosinophils, Week 44, n=1,1,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 25.000 (NA) — Standard deviation could not be calculated for single participant. | 100.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 48, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Eosinophils, Week 48, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | 200.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 52, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Eosinophils, Week 52, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | 300.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 56, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Eosinophils, Week 56, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | 200.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 60, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Eosinophils, Week 60, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | 200.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 64, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Eosinophils, Week 64, n=0,0,1,0 |  |  | 200.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 68, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Eosinophils, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Eosinophils, Week 72, n=0,0,1,0 |  |  | 100.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Eosinophils, Week 76, n=0,0,1,0 |  |  | 100.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Eosinophils, Week 80, n=0,0,1,0 |  |  | 200.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Eosinophils, Week 84, n=0,0,1,0 |  |  | 100.000 (NA) — Standard deviation could not be calculated for single participant. |
  Eosinophils, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Eosinophils, Week 88, n=0,0,1,0 |  |  | 100.000 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 2, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Hematocrit, Week 2, n=10,11,12,2 | 0.587 (6.3505) | 1.183 (4.5122) | -0.387 (4.2431) | -1.480 (3.9739)
  Hematocrit, Week 3, n=9,11,12,2: number analyzed (Participants) | 9 | 11 | 12 | 2
  Hematocrit, Week 3, n=9,11,12,2 | -1.006 (3.4842) | 1.595 (4.8860) | 0.138 (4.7403) | -4.355 (16.3412)
  Hematocrit, Week 4, n=9,11,11,2: number analyzed (Participants) | 9 | 11 | 11 | 2
  Hematocrit, Week 4, n=9,11,11,2 | 0.593 (3.8149) | 0.292 (4.1522) | -1.677 (5.4977) | -7.650 (13.4633)
  Hematocrit, Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Hematocrit, Week 5, n=10,11,10,1 | -1.018 (4.1817) | -1.864 (7.0759) | -0.131 (3.8130) | 4.270 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Hematocrit, Week 8, n=9,10,10,1 | 0.604 (5.0812) | -0.771 (6.0100) | -0.511 (5.3238) | 8.270 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 12, n=6,10,7,1: number analyzed (Participants) | 6 | 10 | 7 | 1
  Hematocrit, Week 12, n=6,10,7,1 | 1.648 (5.3385) | -2.580 (5.8249) | -18.046 (31.9934) | 1.600 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 16, n=7,8,4,1: number analyzed (Participants) | 7 | 8 | 4 | 1
  Hematocrit, Week 16, n=7,8,4,1 | -1.459 (5.9511) | -3.929 (6.5991) | -9.515 (9.0652) | 1.330 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Hematocrit, Week 20, n=5,6,4,1 | 2.638 (6.8653) | -2.392 (7.0021) | -7.138 (7.7051) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Hematocrit, Week 24, n=5,5,3,1 | 0.662 (8.0118) | -2.974 (8.6014) | -7.580 (7.0381) | 2.130 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Hematocrit, Week 28, n=5,3,3,1 | 2.004 (5.2368) | -9.047 (17.3470) | -7.793 (10.5539) | 3.470 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Hematocrit, Week 32, n=4,3,3,1 | 0.365 (9.8402) | -1.917 (4.8321) | -7.827 (12.0475) | -2.930 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Hematocrit, Week 36, n=3,1,3,1 | 1.320 (8.9495) | -16.070 (NA) — Standard deviation could not be calculated for single participant. | -3.420 (4.1589) | -8.800 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Hematocrit, Week 40, n=1,2,2,1 | -4.780 (NA) — Standard deviation could not be calculated for single participant. | -7.755 (11.3632) | -21.690 (14.8068) | -10.130 (NA) — Standard deviation could not be calculated for single participant.
  Hematocrit, Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Hematocrit, Week 44, n=1,2,2,0 | -4.070 (NA) — Standard deviation could not be calculated for single participant. | -1.650 (9.8146) | -8.725 (8.2944) |
  Hematocrit, Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hematocrit, Week 48, n=1,1,1,0 | -4.070 (NA) — Standard deviation could not be calculated for single participant. | 4.180 (NA) — Standard deviation could not be calculated for single participant. | -13.510 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hematocrit, Week 52, n=1,1,1,0 | -8.370 (NA) — Standard deviation could not be calculated for single participant. | -0.840 (NA) — Standard deviation could not be calculated for single participant. | -15.540 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hematocrit, Week 56, n=1,1,1,0 | -12.200 (NA) — Standard deviation could not be calculated for single participant. | 3.060 (NA) — Standard deviation could not be calculated for single participant. | -18.920 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hematocrit, Week 60, n=1,1,1,0 | -7.420 (NA) — Standard deviation could not be calculated for single participant. | 2.230 (NA) — Standard deviation could not be calculated for single participant. | -18.920 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hematocrit, Week 64, n=1,1,1,0 | -5.500 (NA) — Standard deviation could not be calculated for single participant. | -1.950 (NA) — Standard deviation could not be calculated for single participant. | -22.970 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Hematocrit, Week 68, n=1,0,1,0 | -4.310 (NA) — Standard deviation could not be calculated for single participant. |  | -10.810 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hematocrit, Week 72, n=0,0,1,0 |  |  | -12.160 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hematocrit, Week 76, n=0,0,1,0 |  |  | -11.080 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hematocrit, Week 80, n=0,0,1,0 |  |  | -5.680 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hematocrit, Week 84, n=0,0,1,0 |  |  | 1.890 (NA) — Standard deviation could not be calculated for single participant. |
  Hematocrit, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hematocrit, Week 88, n=0,0,1,0 |  |  | -4.320 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 2, n=11,11,12,2 | 1.513 (6.4384) | 1.831 (4.2681) | 0.216 (4.9536) | 2.800 (3.9598)
  Hemoglobin, Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Hemoglobin, Week 3, n=10,11,12,2 | -1.144 (3.3900) | 1.874 (5.1494) | -1.001 (4.4522) | -1.760 (11.5400)
  Hemoglobin, Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Hemoglobin, Week 4, n=10,11,11,2 | 0.821 (3.7955) | 0.564 (3.8663) | -1.301 (5.4112) | -6.225 (11.0662)
  Hemoglobin, Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Hemoglobin, Week 5, n=10,11,10,1 | -0.755 (4.7629) | -2.550 (6.7380) | 0.889 (4.4094) | 2.400 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Hemoglobin, Week 8, n=9,10,10,1 | -0.313 (4.4329) | -1.203 (5.3379) | -0.633 (5.7100) | 8.800 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  Hemoglobin, Week 12, n=7,10,7,1 | -0.121 (6.0781) | -3.316 (5.0843) | -4.847 (7.8349) | 0.800 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Hemoglobin, Week 16, n=8,8,4,1 | -4.005 (8.7693) | -4.451 (6.7484) | -12.315 (9.9652) | 2.400 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Hemoglobin, Week 20, n=5,6,4,1 | 2.906 (8.7982) | -2.668 (7.5665) | -9.055 (9.7215) | 1.600 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Hemoglobin, Week 24, n=5,5,3,1 | 2.148 (8.8710) | -4.124 (8.6379) | -10.137 (7.6478) | 2.400 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Hemoglobin, Week 28, n=5,3,3,1 | 2.410 (6.9580) | -8.843 (21.8918) | -11.723 (11.7348) | 4.800 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Hemoglobin, Week 32, n=4,3,3,1 | 2.838 (11.6934) | -3.430 (6.2333) | -11.350 (15.5425) | -4.000 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Hemoglobin, Week 36, n=3,1,3,1 | 4.303 (8.7527) | -22.030 (NA) — Standard deviation could not be calculated for single participant. | -5.893 (4.9326) | -12.800 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Hemoglobin, Week 40, n=1,2,2,1 | -1.430 (NA) — Standard deviation could not be calculated for single participant. | -7.165 (12.6360) | -24.305 (17.7979) | -11.200 (NA) — Standard deviation could not be calculated for single participant.
  Hemoglobin, Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Hemoglobin, Week 44, n=1,2,2,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -2.815 (13.9936) | -11.970 (12.0491) |
  Hemoglobin, Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hemoglobin, Week 48, n=1,1,1,0 | -2.140 (NA) — Standard deviation could not be calculated for single participant. | 5.310 (NA) — Standard deviation could not be calculated for single participant. | -17.210 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hemoglobin, Week 52, n=1,1,1,0 | -5.710 (NA) — Standard deviation could not be calculated for single participant. | 2.650 (NA) — Standard deviation could not be calculated for single participant. | -18.030 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hemoglobin, Week 56, n=1,1,1,0 | -10.000 (NA) — Standard deviation could not be calculated for single participant. | 6.190 (NA) — Standard deviation could not be calculated for single participant. | -22.130 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hemoglobin, Week 60, n=1,1,1,0 | -5.710 (NA) — Standard deviation could not be calculated for single participant. | 4.420 (NA) — Standard deviation could not be calculated for single participant. | -22.130 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Hemoglobin, Week 64, n=1,1,1,0 | -2.860 (NA) — Standard deviation could not be calculated for single participant. | 3.540 (NA) — Standard deviation could not be calculated for single participant. | -27.870 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Hemoglobin, Week 68, n=1,0,1,0 | -2.140 (NA) — Standard deviation could not be calculated for single participant. |  | -15.570 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hemoglobin, Week 72, n=0,0,1,0 |  |  | -13.110 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hemoglobin, Week 76, n=0,0,1,0 |  |  | -13.110 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hemoglobin, Week 80, n=0,0,1,0 |  |  | -6.560 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hemoglobin, Week 84, n=0,0,1,0 |  |  | 2.460 (NA) — Standard deviation could not be calculated for single participant. |
  Hemoglobin, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hemoglobin, Week 88, n=0,0,1,0 |  |  | -4.100 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 2, n=10,9,9,2: number analyzed (Participants) | 10 | 9 | 9 | 2
  Lymphocytes, Week 2, n=10,9,9,2 | 13.128 (26.4961) | 10.492 (24.1299) | 6.557 (14.9900) | -1.110 (1.5698)
  Lymphocytes, Week 3, n=9,9,11,2: number analyzed (Participants) | 9 | 9 | 11 | 2
  Lymphocytes, Week 3, n=9,9,11,2 | 12.964 (21.6078) | 13.431 (42.8448) | -1.674 (23.4467) | -26.515 (13.9229)
  Lymphocytes, Week 4, n=9,9,9,2: number analyzed (Participants) | 9 | 9 | 9 | 2
  Lymphocytes, Week 4, n=9,9,9,2 | 7.117 (28.8484) | 8.342 (24.6388) | -10.698 (14.0883) | -11.665 (16.4968)
  Lymphocytes, Week 5, n=8,7,9,1: number analyzed (Participants) | 8 | 7 | 9 | 1
  Lymphocytes, Week 5, n=8,7,9,1 | 8.680 (20.3405) | 1.481 (24.0919) | -6.918 (18.1022) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 8, n=7,8,8,1: number analyzed (Participants) | 7 | 8 | 8 | 1
  Lymphocytes, Week 8, n=7,8,8,1 | 2.766 (29.3215) | -0.436 (14.5663) | -0.731 (14.9131) | 36.360 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 12, n=5,7,7,1: number analyzed (Participants) | 5 | 7 | 7 | 1
  Lymphocytes, Week 12, n=5,7,7,1 | 4.374 (31.7985) | 4.237 (25.5117) | -5.857 (18.8992) | -18.180 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 16, n=6,5,4,1: number analyzed (Participants) | 6 | 5 | 4 | 1
  Lymphocytes, Week 16, n=6,5,4,1 | 5.980 (34.3145) | -3.418 (17.2124) | -14.440 (22.8645) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 20, n=4,5,4,1: number analyzed (Participants) | 4 | 5 | 4 | 1
  Lymphocytes, Week 20, n=4,5,4,1 | 7.935 (23.3030) | 4.286 (38.4387) | -22.278 (28.4912) | 9.090 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 24, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Lymphocytes, Week 24, n=4,3,3,1 | 10.143 (32.9329) | 6.063 (42.7487) | -10.130 (24.8888) | 27.270 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 28, n=4,2,3,1: number analyzed (Participants) | 4 | 2 | 3 | 1
  Lymphocytes, Week 28, n=4,2,3,1 | 7.328 (15.4134) | -37.780 (25.1447) | -7.750 (22.4674) | 36.360 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 32, n=3,2,3,1: number analyzed (Participants) | 3 | 2 | 3 | 1
  Lymphocytes, Week 32, n=3,2,3,1 | -1.597 (30.4679) | -8.485 (16.2847) | -12.510 (27.7148) | 27.270 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Lymphocytes, Week 36, n=3,1,3,1 | 18.913 (32.5921) | -24.240 (NA) — Standard deviation could not be calculated for single participant. | -2.037 (17.6391) | 9.090 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 40, n=1,1,2,1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Lymphocytes, Week 40, n=1,1,2,1 | 33.330 (NA) — Standard deviation could not be calculated for single participant. | -30.300 (NA) — Standard deviation could not be calculated for single participant. | -27.855 (11.1086) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Lymphocytes, Week 44, n=1,1,2,0: number analyzed (Participants) | 1 | 1 | 2 | 0
  Lymphocytes, Week 44, n=1,1,2,0 | -8.330 (NA) — Standard deviation could not be calculated for single participant. | -16.670 (NA) — Standard deviation could not be calculated for single participant. | -15.715 (8.0822) |
  Lymphocytes, Week 48, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Lymphocytes, Week 48, n=1,0,1,0 | 8.330 (NA) — Standard deviation could not be calculated for single participant. |  | -21.430 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 52, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Lymphocytes, Week 52, n=1,0,1,0 | 8.330 (NA) — Standard deviation could not be calculated for single participant. |  | -21.430 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 56, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Lymphocytes, Week 56, n=1,0,1,0 | -16.670 (NA) — Standard deviation could not be calculated for single participant. |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 60, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Lymphocytes, Week 60, n=1,0,1,0 | 83.330 (NA) — Standard deviation could not be calculated for single participant. |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 64, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 64, n=0,0,1,0 |  |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 68, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 68, n=0,0,1,0 |  |  | -35.710 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 72, n=0,0,1,0 |  |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 76, n=0,0,1,0 |  |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 80, n=0,0,1,0 |  |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 84, n=0,0,1,0 |  |  | -21.430 (NA) — Standard deviation could not be calculated for single participant. |
  Lymphocytes, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Lymphocytes, Week 88, n=0,0,1,0 |  |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 2, n= 11,11,12,2 | 0.360 (1.0203) | -0.477 (0.5538) | 85.741 (294.1068) | 1.020 (0.9334)
  MCH, Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  MCH, Week 3, n=10,11,12,2 | -0.341 (1.7584) | -1.000 (1.2030) | 15.582 (56.4264) | -0.310 (1.4566)
  MCH, Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  MCH, Week 4, n=10,11,11,2 | 0.042 (1.3267) | -0.942 (1.2281) | -0.277 (2.0468) | -0.735 (1.5203)
  MCH, Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  MCH, Week 5, n=10,11,10,1 | -0.171 (1.5524) | -1.856 (1.4255) | 0.395 (1.8147) | -0.670 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  MCH, Week 8, n=9,10,10,1 | -1.582 (2.0961) | 18.355 (64.3175) | -1.095 (2.1396) | -0.340 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  MCH, Week 12, n=7,10,7,1 | -1.779 (0.8758) | -2.970 (2.2530) | -3.199 (3.6432) | -2.680 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  MCH, Week 16, n=8,8,4,1 | -2.315 (2.6806) | -2.759 (2.4800) | -6.200 (3.1007) | -1.680 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  MCH, Week 20, n=5,6,4,1 | -1.384 (3.1912) | -3.355 (3.6335) | -1.515 (3.7408) | -2.010 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  MCH, Week 24, n=5,5,3,1 | -0.228 (4.4495) | -4.376 (4.3285) | -6.213 (2.3011) | -4.360 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  MCH, Week 28, n=5,3,3,1 | -0.074 (4.0385) | -2.653 (6.3945) | -7.543 (4.5062) | -2.350 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  MCH, Week 32, n=4,3,3,1 | 1.873 (4.2547) | -2.137 (4.9163) | -7.767 (5.6425) | -3.020 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  MCH, Week 36, n=3,1,3,1 | 2.693 (2.3328) | -6.350 (NA) — Standard deviation could not be calculated for single participant. | -5.237 (1.9581) | -8.390 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  MCH, Week 40, n=1,2,2,1 | 3.380 (NA) — Standard deviation could not be calculated for single participant. | -0.255 (2.4819) | -7.705 (3.3870) | -9.060 (NA) — Standard deviation could not be calculated for single participant.
  MCH, Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  MCH, Week 44, n=1,2,2,0 | 4.000 (NA) — Standard deviation could not be calculated for single participant. | -0.710 (0.0566) | -4.425 (1.8314) |
  MCH, Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCH, Week 48, n=1,1,1,0 | 2.150 (NA) — Standard deviation could not be calculated for single participant. | -0.750 (NA) — Standard deviation could not be calculated for single participant. | -5.720 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCH, Week 52, n=1,1,1,0 | 2.150 (NA) — Standard deviation could not be calculated for single participant. | 1.500 (NA) — Standard deviation could not be calculated for single participant. | -6.060 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCH, Week 56, n=1,1,1,0 | -0.620 (NA) — Standard deviation could not be calculated for single participant. | -0.380 (NA) — Standard deviation could not be calculated for single participant. | -4.380 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCH, Week 60, n=1,1,1,0 | 1.230 (NA) — Standard deviation could not be calculated for single participant. | 1.130 (NA) — Standard deviation could not be calculated for single participant. | -4.380 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCH, Week 64, n=1,1,1,0 | 0.920 (NA) — Standard deviation could not be calculated for single participant. | 2.630 (NA) — Standard deviation could not be calculated for single participant. | -10.100 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  MCH, Week 68, n=1,0,1,0 | 0.620 (NA) — Standard deviation could not be calculated for single participant. |  | -5.390 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCH, Week 72, n=0,0,1,0 |  |  | -4.710 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCH, Week 76, n=0,0,1,0 |  |  | -2.360 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCH, Week 80, n=0,0,1,0 |  |  | 0.340 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCH, Week 84, n=0,0,1,0 |  |  | -1.010 (NA) — Standard deviation could not be calculated for single participant. |
  MCH, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCH, Week 88, n=0,0,1,0 |  |  | 1.680 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 2, n= 11,11,12,2 | -0.425 (1.5619) | -0.915 (1.9177) | 0.101 (2.0574) | -2.500 (1.9516)
  MCV, Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  MCV, Week 3, n=10,11,12,2 | -0.735 (1.7112) | -1.025 (2.1801) | 0.158 (1.9350) | -2.940 (4.1578)
  MCV, Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  MCV, Week 4, n=10,11,11,2 | -0.376 (1.5149) | -0.868 (1.6593) | -0.749 (1.7087) | -2.100 (4.5538)
  MCV, Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  MCV, Week 5, n=10,11,10,1 | -0.633 (1.8430) | -0.936 (1.6268) | -0.584 (1.4207) | 1.120 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  MCV, Week 8, n=9,10,10,1 | -0.890 (1.7420) | -1.471 (2.3336) | -1.028 (1.2245) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  MCV, Week 12, n=7,10,7,1 | -1.806 (1.5447) | -2.108 (2.4766) | -2.961 (2.6274) | -2.250 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  MCV, Week 16, n=8,8,4,1 | -1.353 (1.5169) | -2.014 (1.5731) | -3.160 (1.6961) | -2.250 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  MCV, Week 20, n=5,6,4,1 | -2.284 (1.5380) | -2.773 (2.6459) | -2.548 (1.4104) | -3.370 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  MCV, Week 24, n=5,5,3,1 | -2.180 (2.5123) | -2.976 (3.1047) | -3.273 (2.1356) | -4.490 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  MCV, Week 28, n=5,3,3,1 | -0.796 (1.9042) | -1.810 (1.9641) | -3.593 (2.6835) | -3.370 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  MCV, Week 32, n=4,3,3,1 | -0.243 (1.0303) | -0.250 (1.0672) | -3.913 (1.5369) | -1.120 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  MCV, Week 36, n=3,1,3,1 | -0.180 (1.3888) | 0.770 (NA) — Standard deviation could not be calculated for single participant. | -2.397 (1.6820) | -4.490 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  MCV, Week 40, n=1,2,2,1 | -0.510 (NA) — Standard deviation could not be calculated for single participant. | -0.820 (1.1597) | -4.245 (1.6051) | -6.740 (NA) — Standard deviation could not be calculated for single participant.
  MCV, Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  MCV, Week 44, n=1,2,2,0 | -0.310 (NA) — Standard deviation could not be calculated for single participant. | 1.075 (4.2073) | -0.895 (3.3022) |
  MCV, Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCV, Week 48, n=1,1,1,0 | 0.410 (NA) — Standard deviation could not be calculated for single participant. | -1.190 (NA) — Standard deviation could not be calculated for single participant. | -1.560 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCV, Week 52, n=1,1,1,0 | -1.130 (NA) — Standard deviation could not be calculated for single participant. | -1.430 (NA) — Standard deviation could not be calculated for single participant. | -3.440 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCV, Week 56, n=1,1,1,0 | -2.990 (NA) — Standard deviation could not be calculated for single participant. | -2.740 (NA) — Standard deviation could not be calculated for single participant. | -0.220 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCV, Week 60, n=1,1,1,0 | -0.720 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -0.220 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  MCV, Week 64, n=1,1,1,0 | -1.850 (NA) — Standard deviation could not be calculated for single participant. | -2.260 (NA) — Standard deviation could not be calculated for single participant. | -3.780 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  MCV, Week 68, n=1,0,1,0 | -1.540 (NA) — Standard deviation could not be calculated for single participant. |  | 0.220 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCV, Week 72, n=0,0,1,0 |  |  | -3.440 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCV, Week 76, n=0,0,1,0 |  |  | 0.110 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCV, Week 80, n=0,0,1,0 |  |  | 1.560 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCV, Week 84, n=0,0,1,0 |  |  | -1.440 (NA) — Standard deviation could not be calculated for single participant. |
  MCV, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  MCV, Week 88, n=0,0,1,0 |  |  | 1.670 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 2, n=10,9,9,2: number analyzed (Participants) | 10 | 9 | 9 | 2
  Monocytes, Week 2, n=10,9,9,2 | 5.541 (34.2863) | 22.173 (60.1911) | -10.849 (24.6931) | -28.025 (16.9352)
  Monocytes, Week 3, n=9,9,11,2: number analyzed (Participants) | 9 | 9 | 11 | 2
  Monocytes, Week 3, n=9,9,11,2 | -0.646 (30.4427) | -0.434 (19.0109) | -12.739 (34.2922) | -28.025 (16.9352)
  Monocytes, Week 4, n=9,9,9,2: number analyzed (Participants) | 9 | 9 | 9 | 2
  Monocytes, Week 4, n=9,9,9,2 | 1.097 (33.5523) | 13.623 (49.8243) | -10.942 (28.2516) | -23.580 (5.0629)
  Monocytes, Week 5, n=8,8,9,1: number analyzed (Participants) | 8 | 8 | 9 | 1
  Monocytes, Week 5, n=8,8,9,1 | -5.118 (33.7156) | 5.200 (56.5226) | 2.906 (43.9084) | -20.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 8, n=7,8,9,1: number analyzed (Participants) | 7 | 8 | 9 | 1
  Monocytes, Week 8, n=7,8,9,1 | 7.991 (26.3341) | 12.321 (53.9449) | -8.621 (36.1243) | -20.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 12, n=5,7,7,1: number analyzed (Participants) | 5 | 7 | 7 | 1
  Monocytes, Week 12, n=5,7,7,1 | 1.710 (23.3573) | 17.299 (46.0764) | -0.061 (34.6523) | -20.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 16, n=6,5,4,1: number analyzed (Participants) | 6 | 5 | 4 | 1
  Monocytes, Week 16, n=6,5,4,1 | 11.403 (40.0796) | 12.852 (51.7225) | 0.638 (19.3854) | -20.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 20, n=4,5,4,1: number analyzed (Participants) | 4 | 5 | 4 | 1
  Monocytes, Week 20, n=4,5,4,1 | 1.918 (37.7552) | -2.744 (20.6555) | -23.258 (8.0211) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 24, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Monocytes, Week 24, n=4,3,3,1 | 10.033 (44.7607) | 30.770 (53.2952) | -20.633 (18.0268) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 28, n=4,2,3,1: number analyzed (Participants) | 4 | 2 | 3 | 1
  Monocytes, Week 28, n=4,2,3,1 | 13.760 (32.3438) | 0.000 (0.0000) | -9.523 (16.4949) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 32, n=3,2,3,1: number analyzed (Participants) | 3 | 2 | 3 | 1
  Monocytes, Week 32, n=3,2,3,1 | 6.360 (48.8989) | 43.845 (90.2905) | -25.397 (22.5044) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Monocytes, Week 36, n=3,1,3,1 | 13.890 (34.6958) | 50.000 (NA) — Standard deviation could not be calculated for single participant. | -14.287 (24.7452) | -20.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 40, n=1,1,2,1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Monocytes, Week 40, n=1,1,2,1 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 134.620 (NA) — Standard deviation could not be calculated for single participant. | -23.810 (13.4633) | -20.000 (NA) — Standard deviation could not be calculated for single participant.
  Monocytes, Week 44, n=1,1,2,0: number analyzed (Participants) | 1 | 1 | 2 | 0
  Monocytes, Week 44, n=1,1,2,0 | -25.000 (NA) — Standard deviation could not be calculated for single participant. | 46.150 (NA) — Standard deviation could not be calculated for single participant. | -14.285 (20.2020) |
  Monocytes, Week 48, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Monocytes, Week 48, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 52, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Monocytes, Week 52, n=1,0,1,0 | -25.000 (NA) — Standard deviation could not be calculated for single participant. |  | -14.290 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 56, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Monocytes, Week 56, n=1,0,1,0 | 25.000 (NA) — Standard deviation could not be calculated for single participant. |  | -14.290 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 60, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Monocytes, Week 60, n=1,0,1,0 | 25.000 (NA) — Standard deviation could not be calculated for single participant. |  | -14.290 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 64, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 64, n=0,0,1,0 |  |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 68, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 68, n=0,0,1,0 |  |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 72, n=0,0,1,0 |  |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 76, n=0,0,1,0 |  |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 80, n=0,0,1,0 |  |  | -28.570 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 84, n=0,0,1,0 |  |  | -14.290 (NA) — Standard deviation could not be calculated for single participant. |
  Monocytes, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes, Week 88, n=0,0,1,0 |  |  | -42.860 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 2, n=11,11,12,2 | 8.585 (15.9118) | 14.016 (19.2876) | 6.250 (13.3852) | 16.390 (18.2434)
  Platelet count, Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Platelet count, Week 3, n=10,11,12,2 | -0.057 (12.3510) | 5.440 (11.6551) | -1.445 (10.3439) | 8.325 (15.3654)
  Platelet count, Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Platelet count, Week 4, n=10,11,11,2 | -0.921 (7.2065) | -4.057 (9.0344) | -8.287 (8.2288) | 11.095 (7.1630)
  Platelet count, Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Platelet count, Week 5, n=10,11,10,1 | -4.600 (8.7256) | 0.846 (24.9856) | -3.811 (11.4610) | 18.180 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Platelet count, Week 8, n=9,10,10,1 | 2.416 (12.6516) | 2.883 (9.9460) | 2.206 (11.3950) | 18.690 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 12, n=7, 9,7,1: number analyzed (Participants) | 7 | 9 | 7 | 1
  Platelet count, Week 12, n=7, 9,7,1 | 6.046 (15.8538) | -3.291 (9.0120) | -1.393 (12.3185) | 9.090 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Platelet count, Week 16, n=8,8,4,1 | 7.735 (21.7273) | -7.453 (10.0630) | 2.405 (29.4379) | 14.650 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Platelet count, Week 20, n=5,6,4,1 | -3.764 (11.6336) | -5.373 (11.3944) | 2.958 (22.8724) | 14.140 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Platelet count, Week 24, n=5,5,3,1 | 0.846 (18.2657) | 5.036 (21.6048) | -0.247 (28.6042) | 23.740 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Platelet count, Week 28, n=5,3,3,1 | -1.656 (13.0916) | -5.473 (16.0800) | -7.450 (17.5451) | 17.680 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Platelet count, Week 32, n=4,3,3,1 | -20.275 (52.6390) | -8.827 (11.3729) | 0.790 (28.4249) | 39.900 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Platelet count, Week 36, n=3,1,3,1 | -2.597 (19.7730) | -8.820 (NA) — Standard deviation could not be calculated for single participant. | 2.967 (18.8553) | 50.000 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Platelet count, Week 40, n=1,2,2,1 | 9.630 (NA) — Standard deviation could not be calculated for single participant. | 0.785 (4.2356) | -3.070 (23.6315) | 57.580 (NA) — Standard deviation could not be calculated for single participant.
  Platelet count, Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Platelet count, Week 44, n=1,2,2,0 | 0.460 (NA) — Standard deviation could not be calculated for single participant. | -25.160 (36.1756) | -9.450 (9.8571) |
  Platelet count, Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Platelet count, Week 48, n=1,1,1,0 | -5.960 (NA) — Standard deviation could not be calculated for single participant. | -1.680 (NA) — Standard deviation could not be calculated for single participant. | -8.680 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Platelet count, Week 52, n=1,1,1,0 | -2.750 (NA) — Standard deviation could not be calculated for single participant. | -10.080 (NA) — Standard deviation could not be calculated for single participant. | -1.650 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Platelet count, Week 56, n=1,1,1,0 | 0.920 (NA) — Standard deviation could not be calculated for single participant. | 7.140 (NA) — Standard deviation could not be calculated for single participant. | -7.440 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Platelet count, Week 60, n=1,1,1,0 | 16.060 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -7.440 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Platelet count, Week 64, n=1,1,1,0 | -7.340 (NA) — Standard deviation could not be calculated for single participant. | -7.140 (NA) — Standard deviation could not be calculated for single participant. | -3.310 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Platelet count, Week 68, n=1,0,1,0 | -0.460 (NA) — Standard deviation could not be calculated for single participant. |  | -11.570 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Platelet count, Week 72, n=0,0,1,0 |  |  | -2.070 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Platelet count, Week 76, n=0,0,1,0 |  |  | -26.860 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Platelet count, Week 80, n=0,0,1,0 |  |  | -16.120 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Platelet count, Week 84, n=0,0,1,0 |  |  | -16.120 (NA) — Standard deviation could not be calculated for single participant. |
  Platelet count, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Platelet count, Week 88, n=0,0,1,0 |  |  | -31.400 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 2, n= 10,9,9,2: number analyzed (Participants) | 10 | 9 | 9 | 2
  Total Neutrophils, Week 2, n= 10,9,9,2 | 6.689 (45.0555) | -6.798 (37.2810) | -3.907 (19.8441) | 0.380 (0.5374)
  Total Neutrophils, Week 3, n=9,9,11,2: number analyzed (Participants) | 9 | 9 | 11 | 2
  Total Neutrophils, Week 3, n=9,9,11,2 | -1.933 (38.2961) | -9.604 (34.8399) | -1.496 (28.6849) | 13.885 (25.0245)
  Total Neutrophils, Week 4, n=9,9,9,2: number analyzed (Participants) | 9 | 9 | 9 | 2
  Total Neutrophils, Week 4, n=9,9,9,2 | -0.562 (48.2259) | 10.019 (70.2338) | -17.251 (23.9291) | -14.600 (5.7558)
  Total Neutrophils, Week 5, n=8,8,9,1: number analyzed (Participants) | 8 | 8 | 9 | 1
  Total Neutrophils, Week 5, n=8,8,9,1 | -14.485 (23.6250) | -10.721 (27.2234) | -3.097 (38.5928) | 36.840 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 8, n=7,8,9,1: number analyzed (Participants) | 7 | 8 | 9 | 1
  Total Neutrophils, Week 8, n=7,8,9,1 | -6.409 (22.6409) | -8.959 (32.9931) | -6.433 (31.7619) | 47.370 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 12, n=5,7,7,1: number analyzed (Participants) | 5 | 7 | 7 | 1
  Total Neutrophils, Week 12, n=5,7,7,1 | -7.292 (29.7757) | -4.930 (24.9495) | -0.051 (28.1875) | 36.840 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 16, n=6,5,4,1: number analyzed (Participants) | 6 | 5 | 4 | 1
  Total Neutrophils, Week 16, n=6,5,4,1 | -11.992 (26.9160) | -17.300 (32.1449) | -11.233 (29.4360) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 20, n=4,5,4,1: number analyzed (Participants) | 4 | 5 | 4 | 1
  Total Neutrophils, Week 20, n=4,5,4,1 | -8.668 (40.6758) | -22.398 (33.4115) | -37.638 (14.2156) | 31.580 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 24, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Total Neutrophils, Week 24, n=4,3,3,1 | -9.695 (39.8258) | 537.517 (875.0638) | -25.860 (19.3876) | 31.580 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 28, n=4,1,3,1: number analyzed (Participants) | 4 | 1 | 3 | 1
  Total Neutrophils, Week 28, n=4,1,3,1 | -4.173 (38.7614) | -23.910 (NA) — Standard deviation could not be calculated for single participant. | -15.737 (30.5955) | -5.260 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 32, n=3,2,3,1: number analyzed (Participants) | 3 | 2 | 3 | 1
  Total Neutrophils, Week 32, n=3,2,3,1 | -17.917 (30.8176) | 43.785 (117.2595) | -27.140 (12.5575) | 68.420 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Total Neutrophils, Week 36, n=3,1,3,1 | -19.807 (28.6365) | -13.120 (NA) — Standard deviation could not be calculated for single participant. | -22.173 (19.2353) | 47.370 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 40, n=1,1,2,1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Total Neutrophils, Week 40, n=1,1,2,1 | 23.810 (NA) — Standard deviation could not be calculated for single participant. | 57.920 (NA) — Standard deviation could not be calculated for single participant. | -18.750 (26.5165) | -5.260 (NA) — Standard deviation could not be calculated for single participant.
  Total Neutrophils, Week 44, n=1,1,2,0: number analyzed (Participants) | 1 | 1 | 2 | 0
  Total Neutrophils, Week 44, n=1,1,2,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 1.810 (NA) — Standard deviation could not be calculated for single participant. | -15.130 (13.9583) |
  Total Neutrophils, Week 48, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Total Neutrophils, Week 48, n=1,0,1,0 | -14.290 (NA) — Standard deviation could not be calculated for single participant. |  | -23.680 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 52, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Total Neutrophils, Week 52, n=1,0,1,0 | 61.900 (NA) — Standard deviation could not be calculated for single participant. |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 56, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Total Neutrophils, Week 56, n=1,0,1,0 | 4.760 (NA) — Standard deviation could not be calculated for single participant. |  | -21.050 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 60, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Total Neutrophils, Week 60, n=1,0,1,0 | 33.330 (NA) — Standard deviation could not be calculated for single participant. |  | -21.050 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 64, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 64, n=0,0,1,0 |  |  | -13.160 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 68, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 68, n=0,0,1,0 |  |  | -15.790 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 72, n=0,0,1,0 |  |  | -21.050 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 76, n=0,0,1,0 |  |  | -39.470 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 80, n=0,0,1,0 |  |  | -15.790 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 84, n=0,0,1,0 |  |  | -21.050 (NA) — Standard deviation could not be calculated for single participant. |
  Total Neutrophils, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total Neutrophils, Week 88, n=0,0,1,0 |  |  | -28.950 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 2, n=11,11,12,2 | 6.813 (29.4392) | -2.077 (26.5166) | 0.445 (15.7801) | -2.220 (0.7920)
  WBC count, Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  WBC count, Week 3, n=10,11,12,2 | 1.486 (24.4918) | -2.625 (26.9770) | -3.928 (20.8967) | -1.715 (6.3569)
  WBC count, Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  WBC count, Week 4, n=10,11,11,2 | -0.001 (28.4127) | 5.575 (51.6285) | -12.681 (18.5282) | -12.505 (9.8217)
  WBC count, Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  WBC count, Week 5, n=10,11,10,1 | -4.419 (20.0450) | -10.823 (16.8580) | -3.190 (31.2346) | 19.440 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  WBC count, Week 8, n=9,10,10,1 | -3.917 (18.3295) | -8.811 (23.2822) | -2.931 (23.8804) | 30.560 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  WBC count, Week 12, n=7,10,7,1 | -1.723 (19.0232) | -10.782 (18.8356) | 2.471 (25.2046) | 8.330 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  WBC count, Week 16, n=8,8,4,1 | -4.974 (23.1270) | -16.450 (20.2532) | -11.380 (20.6158) | -2.780 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  WBC count, Week 20, n=5,6,4,1 | -3.674 (25.9508) | -15.540 (21.0813) | -30.808 (10.3805) | 19.440 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  WBC count, Week 24, n=5,5,3,1 | -0.176 (33.0932) | 2.760 (47.1809) | -23.037 (13.3905) | 27.780 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  WBC count, Week 28, n=5,3,3,1 | 3.036 (22.6756) | -10.843 (8.9673) | -15.997 (15.6148) | 8.330 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  WBC count, Week 32, n=4,3,3,1 | -9.978 (22.7259) | 14.077 (73.8998) | -24.583 (11.4453) | 47.220 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  WBC count, Week 36, n=3,1,3,1 | -6.547 (29.9390) | -8.810 (NA) — Standard deviation could not be calculated for single participant. | -17.613 (6.2673) | 27.780 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  WBC count, Week 40, n=1,2,2,1 | 23.080 (NA) — Standard deviation could not be calculated for single participant. | 21.725 (36.8756) | -22.375 (12.3532) | -5.560 (NA) — Standard deviation could not be calculated for single participant.
  WBC count, Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  WBC count, Week 44, n=1,2,2,0 | -7.690 (NA) — Standard deviation could not be calculated for single participant. | -2.525 (6.6822) | -17.225 (0.7849) |
  WBC count, Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  WBC count, Week 48, n=1,1,1,0 | -5.130 (NA) — Standard deviation could not be calculated for single participant. | -18.840 (NA) — Standard deviation could not be calculated for single participant. | -25.760 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  WBC count, Week 52, n=1,1,1,0 | 35.900 (NA) — Standard deviation could not be calculated for single participant. | -8.700 (NA) — Standard deviation could not be calculated for single participant. | -9.090 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  WBC count, Week 56, n=1,1,1,0 | -7.690 (NA) — Standard deviation could not be calculated for single participant. | -2.900 (NA) — Standard deviation could not be calculated for single participant. | -25.760 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  WBC count, Week 60, n=1,1,1,0 | 43.590 (NA) — Standard deviation could not be calculated for single participant. | -10.140 (NA) — Standard deviation could not be calculated for single participant. | -25.760 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  WBC count, Week 64, n=1,1,1,0 | 15.380 (NA) — Standard deviation could not be calculated for single participant. | -7.250 (NA) — Standard deviation could not be calculated for single participant. | -24.240 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  WBC count, Week 68, n=1,0,1,0 | -2.560 (NA) — Standard deviation could not be calculated for single participant. |  | -25.760 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC count, Week 72, n=0,0,1,0 |  |  | -27.270 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC count, Week 76, n=0,0,1,0 |  |  | -42.420 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC count, Week 80, n=0,0,1,0 |  |  | -27.270 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC count, Week 84, n=0,0,1,0 |  |  | -24.240 (NA) — Standard deviation could not be calculated for single participant. |
  WBC count, Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  WBC count, Week 88, n=0,0,1,0 |  |  | -36.360 (NA) — Standard deviation could not be calculated for single participant. |

5. Primary Outcome: Percent Change From Baseline in Hematology Parameters During Combination Treatment Period: International Normalized Ratio (INR), Prothrombin Time (PT), Partial Thromboplastin Time (PTT)
Description: Blood samples were collected to analyze the hematology parameters: INR, PT and PTT. Baseline value is the latest GSK2636771 pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100 multiplied by (post-Baseline visit value minus Baseline divided by Baseline).
Time Frame: Baseline (Day 1), Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 10 | 9 | 11 | 1
Percent change
  INR, n=9,9,11,1: number analyzed (Participants) | 9 | 9 | 11 | 1
  INR, n=9,9,11,1 | -9.266 (31.1026) | 1.230 (3.7353) | 0.287 (0.6848) | 11.110 (NA) — Standard deviation could not be calculated for single participant.
  PT, n=9,9,11,0: number analyzed (Participants) | 9 | 9 | 11 | 0
  PT, n=9,9,11,0 | 114.626 (344.5226) | -0.677 (5.5257) | 1.328 (1.9928) |
  PTT, n=10,9,11,0: number analyzed (Participants) | 10 | 9 | 11 | 0
  PTT, n=10,9,11,0 | 252.137 (799.4078) | 3.480 (11.0842) | 4.596 (4.3461) |

6. Primary Outcome: Percent Change From Baseline in Chemistry Parameters in Combination Treatment Period:ALT, Albumin, ALP, AST, Calcium, CO2, Chloride, Creatinine, Direct Bilirubin, Glucose, Lactate Dehydrogenase, Magnesium, Potassium, Sodium, Total Bilirubin, Total Protein
Description: Blood samples were collected to analyze the chemistry parameters: ALT, Albumin, Alkaline phosphatase (ALP), Aspartate amino transferase (AST), Calcium, Carbon dioxide (CO2), Chloride, Creatinine, Direct bilirubin, Glucose, Lactate dehydrogenase, Magnesium, Potassium, Sodium, Total bilirubin and Total protein. Baseline value is the latest GSK2636771 pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100 multiplied by (post-Baseline visit value minus Baseline divided by Baseline).
Time Frame: Baseline (Day 1), Weeks 1,2,3,4,5,8,12,16,20,24,28,32,36,40,44,48,52,56,60,64,68,72,76,80,84 and 88
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Percent change
  ALT:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  ALT:Week 1, n=0,0,3,1 |  |  | 19.283 (22.1495) | 42.860 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 2, n=11,11,12,2 | 24.745 (33.0344) | 26.454 (40.8793) | 37.503 (19.7223) | 35.715 (10.1046)
  ALT:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  ALT:Week 3, n=10,11,12,2 | 23.264 (31.2843) | 32.356 (43.4898) | 30.123 (16.5230) | 14.285 (20.2020)
  ALT:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  ALT:Week 4, n=10,11,11,2 | 29.468 (30.6030) | 42.434 (57.8048) | 58.457 (62.8020) | 28.575 (20.2020)
  ALT:Week 5, n= 10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  ALT:Week 5, n= 10,11,10,1 | 29.714 (30.3371) | 45.801 (36.5261) | 39.647 (33.2853) | 28.570 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  ALT:Week 8, n=9,10,10,1 | 53.636 (62.0500) | 57.566 (61.0093) | 32.372 (26.1619) | 14.290 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  ALT:Week 12, n=7,10,7,1 | 31.460 (37.8221) | 45.549 (37.9079) | 21.621 (22.5414) | 28.570 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  ALT:Week 16, n=8,8,4,1 | 30.841 (36.3547) | 37.271 (41.2228) | 25.113 (50.7297) | 57.140 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  ALT:Week 20, n=5,6,4,1 | 31.442 (28.4784) | 17.172 (47.1226) | 19.048 (26.0889) | 42.860 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  ALT:Week 24, n=5,5,3,1 | 25.280 (29.7220) | 23.628 (56.9181) | 26.863 (9.1878) | 57.140 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  ALT:Week 28, n=5,4,3,1 | 48.140 (25.3878) | -15.128 (35.7843) | 9.793 (10.6010) | 57.140 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  ALT:Week 32, n=4,3,3,1 | 44.170 (29.4179) | -31.510 (5.3476) | 7.970 (11.6457) | 42.860 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  ALT:Week 36, n=3,1,3,1 | 53.580 (26.3536) | -6.670 (NA) — Standard deviation could not be calculated for single participant. | 3.180 (11.3589) | -14.290 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  ALT:Week 40, n=1,2,2,1 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -27.060 (0.5515) | -0.495 (8.1388) | 14.290 (NA) — Standard deviation could not be calculated for single participant.
  ALT:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  ALT:Week 44, n=1,2,2,0 | 50.000 (NA) — Standard deviation could not be calculated for single participant. | 6.075 (66.8287) | -3.125 (4.4194) |
  ALT:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALT:Week 48, n=1,1,1,0 | 100.000 (NA) — Standard deviation could not be calculated for single participant. | -19.610 (NA) — Standard deviation could not be calculated for single participant. | 15.790 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALT:Week 52, n=1,1,1,0 | 50.000 (NA) — Standard deviation could not be calculated for single participant. | -43.140 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALT:Week 56, n=1,1,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -47.060 (NA) — Standard deviation could not be calculated for single participant. | -5.260 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALT:Week 60, n=1,1,1,0 | 25.000 (NA) — Standard deviation could not be calculated for single participant. | -33.330 (NA) — Standard deviation could not be calculated for single participant. | 15.790 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALT:Week 64, n=1,1,1,0 | 50.000 (NA) — Standard deviation could not be calculated for single participant. | -49.020 (NA) — Standard deviation could not be calculated for single participant. | 15.790 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALT:Week 68, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | 26.320 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT:Week 72, n=0,0,1,0 |  |  | 42.110 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT:Week 76, n=0,0,1,0 |  |  | -15.790 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT:Week 80, n=0,0,1,0 |  |  | 10.530 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT:Week 84, n=0,0,1,0 |  |  | -5.260 (NA) — Standard deviation could not be calculated for single participant. |
  ALT:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT:Week 88, n=0,0,1,0 |  |  | 5.260 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Albumin:Week 1, n=0,0,3,1 |  |  | 1.450 (2.5115) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 2, n=11,11,12,2 | 1.895 (7.5980) | -2.445 (5.0415) | 0.137 (6.3551) | -3.230 (10.7197)
  Albumin:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Albumin:Week 3, n=10,11,12,2 | 0.642 (7.8696) | -1.401 (5.7148) | -2.284 (11.8853) | -5.670 (11.0874)
  Albumin:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Albumin:Week 4, n=10,11,11,2 | 2.024 (3.2354) | -1.667 (3.7915) | -1.075 (4.8150) | -8.665 (3.0335)
  Albumin:Week 5, n= 10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Albumin:Week 5, n= 10,11,10,1 | 0.625 (5.4575) | -0.532 (4.3994) | 0.597 (5.0133) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Albumin:Week 8, n=9,10,10,1 | 3.182 (3.5152) | -2.282 (3.3157) | 1.648 (6.0048) | 10.870 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 12, n=6,10,7,1: number analyzed (Participants) | 6 | 10 | 7 | 1
  Albumin:Week 12, n=6,10,7,1 | 1.805 (7.7531) | -4.026 (5.6375) | 0.547 (4.3503) | -2.170 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Albumin:Week 16, n=8,8,4,1 | 0.755 (6.1997) | -4.880 (4.0347) | -3.378 (5.6123) | 2.170 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Albumin:Week 20, n=5,6,4,1 | 0.596 (10.1128) | -3.827 (6.8293) | 0.130 (6.2519) | 2.170 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Albumin:Week 24, n=5,5,3,1 | 1.070 (5.9309) | -4.052 (4.0523) | -1.130 (3.9870) | 4.350 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Albumin:Week 28, n=5,4,3,1 | 0.668 (5.4560) | -8.870 (8.1232) | 1.147 (5.8101) | 2.170 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Albumin:Week 32, n=4,3,3,1 | 3.635 (8.4967) | -5.747 (4.0772) | -3.603 (7.9065) | -4.350 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Albumin:Week 36, n=3,1,3,1 | 2.403 (4.6570) | -9.300 (NA) — Standard deviation could not be calculated for single participant. | -1.180 (5.0541) | -2.170 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Albumin:Week 40, n=1,2,2,1 | -9.300 (NA) — Standard deviation could not be calculated for single participant. | -4.650 (9.8712) | -7.730 (4.7800) | 2.170 (NA) — Standard deviation could not be calculated for single participant.
  Albumin:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Albumin:Week 44, n=1,2,2,0 | -4.650 (NA) — Standard deviation could not be calculated for single participant. | -3.490 (4.9356) | -0.905 (10.5005) |
  Albumin:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Albumin:Week 48, n=1,1,1,0 | -4.650 (NA) — Standard deviation could not be calculated for single participant. | 2.330 (NA) — Standard deviation could not be calculated for single participant. | -8.330 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Albumin:Week 52, n=1,1,1,0 | -6.980 (NA) — Standard deviation could not be calculated for single participant. | -6.980 (NA) — Standard deviation could not be calculated for single participant. | -8.330 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Albumin:Week 56, n=1,1,1,0 | -9.300 (NA) — Standard deviation could not be calculated for single participant. | -6.980 (NA) — Standard deviation could not be calculated for single participant. | -8.330 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Albumin:Week 60, n=1,1,1,0 | -9.300 (NA) — Standard deviation could not be calculated for single participant. | -4.650 (NA) — Standard deviation could not be calculated for single participant. | -11.110 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Albumin:Week 64, n=1,1,1,0 | -6.980 (NA) — Standard deviation could not be calculated for single participant. | -2.330 (NA) — Standard deviation could not be calculated for single participant. | -8.330 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Albumin:Week 68, n=1,0,1,0 | -6.980 (NA) — Standard deviation could not be calculated for single participant. |  | -5.560 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Albumin:Week 72, n=0,0,1,0 |  |  | -8.330 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Albumin:Week 76, n=0,0,1,0 |  |  | -11.110 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Albumin:Week 80, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Albumin:Week 84, n=0,0,1,0 |  |  | -2.780 (NA) — Standard deviation could not be calculated for single participant. |
  Albumin:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Albumin:Week 88, n=0,0,1,0 |  |  | -13.890 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  ALP:Week 1, n=0,0,3,1 |  |  | -4.147 (6.3515) | -5.410 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 2, n=11,10,12,2: number analyzed (Participants) | 11 | 10 | 12 | 2
  ALP:Week 2, n=11,10,12,2 | 3.165 (15.9188) | 2.881 (13.4737) | 2.665 (19.2406) | -3.660 (16.4897)
  ALP:Week 3, n=10,10,12,2: number analyzed (Participants) | 10 | 10 | 12 | 2
  ALP:Week 3, n=10,10,12,2 | 6.972 (10.8810) | 5.072 (17.3872) | -0.942 (15.7497) | 10.000 (14.1421)
  ALP:Week 4, n=10,10,11,2: number analyzed (Participants) | 10 | 10 | 11 | 2
  ALP:Week 4, n=10,10,11,2 | 3.496 (11.7663) | 11.790 (21.9785) | -2.819 (16.9420) | 21.665 (16.4968)
  ALP:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  ALP:Week 5, n=10,11,10,1 | 3.251 (14.5791) | 11.901 (20.1563) | 0.269 (17.4773) | 8.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  ALP:Week 8, n=9,10,10,1 | 4.360 (12.8823) | 12.790 (27.1346) | -1.651 (18.0020) | 28.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  ALP:Week 12, n=7,10,7,1 | 1.306 (18.5543) | 11.758 (37.2451) | -3.350 (17.4644) | 6.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  ALP:Week 16, n=8,8,4,1 | 2.364 (35.6322) | 18.066 (54.1061) | -10.875 (7.5274) | 22.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  ALP:Week 20, n=5,6,4,1 | -19.620 (7.2268) | 25.492 (87.1563) | -13.655 (8.0427) | 18.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  ALP:Week 24, n=5,5,3,1 | -20.088 (8.7955) | 71.670 (167.7482) | -18.933 (5.0374) | 16.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  ALP:Week 28, n=5,4,3,1 | -15.240 (11.3616) | 75.765 (161.7779) | -16.040 (11.2100) | 14.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  ALP:Week 32, n=4,3,3,1 | -16.640 (11.5509) | 84.763 (119.3992) | -10.653 (22.0605) | 38.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  ALP:Week 36, n=3,1,3,1 | -9.937 (4.2691) | 173.030 (NA) — Standard deviation could not be calculated for single participant. | -9.480 (18.9095) | 24.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  ALP:Week 40, n=1,2,2,1 | -3.850 (NA) — Standard deviation could not be calculated for single participant. | 24.230 (59.4818) | -20.895 (0.1485) | 12.000 (NA) — Standard deviation could not be calculated for single participant.
  ALP:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  ALP:Week 44, n=1,2,2,0 | 5.770 (NA) — Standard deviation could not be calculated for single participant. | 51.715 (133.4381) | -14.000 (19.7990) |
  ALP:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALP:Week 48, n=1,1,1,0 | 1.920 (NA) — Standard deviation could not be calculated for single participant. | -29.460 (NA) — Standard deviation could not be calculated for single participant. | -21.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALP:Week 52, n=1,1,1,0 | 9.620 (NA) — Standard deviation could not be calculated for single participant. | -44.190 (NA) — Standard deviation could not be calculated for single participant. | -15.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALP:Week 56, n=1,1,1,0 | 1.920 (NA) — Standard deviation could not be calculated for single participant. | -41.090 (NA) — Standard deviation could not be calculated for single participant. | -10.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALP:Week 60, n=1,1,1,0 | -15.380 (NA) — Standard deviation could not be calculated for single participant. | -24.810 (NA) — Standard deviation could not be calculated for single participant. | -8.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  ALP:Week 64, n=1,1,1,0 | -19.230 (NA) — Standard deviation could not be calculated for single participant. | -37.980 (NA) — Standard deviation could not be calculated for single participant. | -11.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  ALP:Week 68, n=1,0,1,0 | -9.620 (NA) — Standard deviation could not be calculated for single participant. |  | -12.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALP:Week 72, n=0,0,1,0 |  |  | -13.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALP:Week 76, n=0,0,1,0 |  |  | -26.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALP:Week 80, n=0,0,1,0 |  |  | -14.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALP:Week 84, n=0,0,1,0 |  |  | -9.000 (NA) — Standard deviation could not be calculated for single participant. |
  ALP:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALP:Week 88, n=0,0,1,0 |  |  | -3.000 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  AST:Week 1, n=0,0,3,1 |  |  | 17.083 (4.0182) | 27.780 (NA) — Standard deviation could not be calculated for single participant.
  AST:Week 2, n=11,11,12,1: number analyzed (Participants) | 11 | 11 | 12 | 1
  AST:Week 2, n=11,11,12,1 | 15.050 (26.7980) | 10.286 (21.5863) | 18.918 (29.8292) | 11.110 (NA) — Standard deviation could not be calculated for single participant.
  AST:Week 3, n=10,11,12,1: number analyzed (Participants) | 10 | 11 | 12 | 1
  AST:Week 3, n=10,11,12,1 | 8.979 (17.9450) | 6.365 (20.9402) | 9.471 (29.6507) | -5.560 (NA) — Standard deviation could not be calculated for single participant.
  AST:Week 4, n=10,11,11,1: number analyzed (Participants) | 10 | 11 | 11 | 1
  AST:Week 4, n=10,11,11,1 | 10.427 (13.4082) | 24.937 (41.2658) | 8.762 (32.5615) | 22.220 (NA) — Standard deviation could not be calculated for single participant.
  AST:Week 5, n=10,11,10,0: number analyzed (Participants) | 10 | 11 | 10 | 0
  AST:Week 5, n=10,11,10,0 | 7.934 (22.4691) | 31.374 (27.5174) | 13.756 (38.8757) |
  AST:Week 8, n=9,10,10,0: number analyzed (Participants) | 9 | 10 | 10 | 0
  AST:Week 8, n=9,10,10,0 | 33.676 (31.1394) | 25.584 (65.6073) | 11.455 (21.3067) |
  AST:Week 12, n=7,10,7,0: number analyzed (Participants) | 7 | 10 | 7 | 0
  AST:Week 12, n=7,10,7,0 | 16.030 (15.7802) | 29.940 (33.2473) | 27.560 (28.1989) |
  AST:Week 16, n=8,8,4,0: number analyzed (Participants) | 8 | 8 | 4 | 0
  AST:Week 16, n=8,8,4,0 | 31.790 (33.3934) | 21.604 (29.1979) | 32.398 (52.6950) |
  AST:Week 20, n=5,6,4,0: number analyzed (Participants) | 5 | 6 | 4 | 0
  AST:Week 20, n=5,6,4,0 | 13.548 (8.4530) | 3.055 (33.4592) | 23.855 (14.8504) |
  AST:Week 24, n=5,5,3,0: number analyzed (Participants) | 5 | 5 | 3 | 0
  AST:Week 24, n=5,5,3,0 | 14.364 (11.9664) | 9.360 (38.6693) | 6.807 (32.9686) |
  AST:Week 28, n=5,4,3,0: number analyzed (Participants) | 5 | 4 | 3 | 0
  AST:Week 28, n=5,4,3,0 | 23.032 (18.8242) | -12.230 (25.1693) | 15.000 (13.2288) |
  AST:Week 32, n=4,3,3,0: number analyzed (Participants) | 4 | 3 | 3 | 0
  AST:Week 32, n=4,3,3,0 | 17.590 (14.7541) | -39.743 (7.1666) | 26.943 (30.4636) |
  AST:Week 36, n=3,1,3,0: number analyzed (Participants) | 3 | 1 | 3 | 0
  AST:Week 36, n=3,1,3,0 | 23.717 (4.7627) | -5.000 (NA) — Standard deviation could not be calculated for single participant. | 13.193 (27.9755) |
  AST:Week 40, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  AST:Week 40, n=1,2,2,0 | 35.290 (NA) — Standard deviation could not be calculated for single participant. | -12.060 (25.3710) | -2.085 (14.7290) |
  AST:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  AST:Week 44, n=1,2,2,0 | 23.530 (NA) — Standard deviation could not be calculated for single participant. | 2.060 (46.5842) | 6.250 (26.5165) |
  AST:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  AST:Week 48, n=1,1,1,0 | 35.290 (NA) — Standard deviation could not be calculated for single participant. | -29.410 (NA) — Standard deviation could not be calculated for single participant. | -18.750 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  AST:Week 52, n=1,1,1,0 | 11.760 (NA) — Standard deviation could not be calculated for single participant. | -50.000 (NA) — Standard deviation could not be calculated for single participant. | -25.000 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  AST:Week 56, n=1,1,1,0 | 17.650 (NA) — Standard deviation could not be calculated for single participant. | -50.000 (NA) — Standard deviation could not be calculated for single participant. | -18.750 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  AST:Week 60, n=1,1,1,0 | 11.760 (NA) — Standard deviation could not be calculated for single participant. | -39.710 (NA) — Standard deviation could not be calculated for single participant. | -12.500 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  AST:Week 64, n=1,1,1,0 | 58.820 (NA) — Standard deviation could not be calculated for single participant. | -57.350 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  AST:Week 68, n=1,0,1,0 | 47.060 (NA) — Standard deviation could not be calculated for single participant. |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  AST:Week 72, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  AST:Week 76, n=0,0,1,0 |  |  | -31.250 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  AST:Week 80, n=0,0,1,0 |  |  | 12.500 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  AST:Week 84, n=0,0,1,0 |  |  | -18.750 (NA) — Standard deviation could not be calculated for single participant. |
  AST:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  AST:Week 88, n=0,0,1,0 |  |  | -18.750 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Calcium:Week 1, n=0,0,3,1 |  |  | -5.307 (1.8287) | -3.530 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 2, n=11,11,12,2 | -4.765 (6.1486) | -3.451 (4.2733) | -8.617 (6.2882) | -5.240 (9.2207)
  Calcium:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Calcium:Week 3, n=10,11,12,2 | -4.547 (7.2916) | -1.819 (3.4578) | -4.798 (3.5578) | -1.830 (7.3963)
  Calcium:Week 4, n=10,10,11,2: number analyzed (Participants) | 10 | 10 | 11 | 2
  Calcium:Week 4, n=10,10,11,2 | -4.768 (5.4864) | -2.178 (5.4456) | -6.373 (4.8535) | -6.960 (13.4492)
  Calcium:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Calcium:Week 5, n=10,11,10,1 | -5.613 (4.6806) | -1.622 (5.5177) | -4.908 (4.6481) | 3.400 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Calcium:Week 8, n=9,10,10,1 | -5.359 (3.8797) | -2.750 (3.5749) | -4.512 (3.8618) | 2.980 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 12, n=6,10,7,1: number analyzed (Participants) | 6 | 10 | 7 | 1
  Calcium:Week 12, n=6,10,7,1 | -3.578 (5.6792) | -2.962 (2.8943) | -6.034 (5.0312) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Calcium:Week 16, n=8,8,4,1 | -4.259 (4.3485) | -4.580 (3.6844) | -6.105 (3.9821) | 1.700 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Calcium:Week 20, n=5,6,4,1 | -5.090 (5.8459) | 0.690 (4.7342) | -5.103 (3.7503) | 1.280 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Calcium:Week 24, n=5,5,3,1 | -3.500 (2.1050) | -2.694 (1.8159) | -5.127 (4.9099) | 5.110 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Calcium:Week 28, n=5,4,3,1 | -2.380 (2.0033) | -3.428 (4.0359) | -5.423 (6.4883) | 5.530 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Calcium:Week 32, n=4,3,3,1 | -4.595 (3.5314) | -0.747 (2.2739) | -6.553 (5.6435) | 1.280 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Calcium:Week 36, n=3,1,3,1 | -5.473 (3.5181) | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -5.210 (5.7373) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 40, n=1,1,2,1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Calcium:Week 40, n=1,1,2,1 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -4.400 (NA) — Standard deviation could not be calculated for single participant. | -8.275 (11.1086) | 2.130 (NA) — Standard deviation could not be calculated for single participant.
  Calcium:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Calcium:Week 44, n=1,2,2,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 2.075 (7.6014) | -1.760 (9.6732) |
  Calcium:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Calcium:Week 48, n=1,1,1,0 | -8.160 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -6.450 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Calcium:Week 52, n=1,1,1,0 | -1.020 (NA) — Standard deviation could not be calculated for single participant. | 2.130 (NA) — Standard deviation could not be calculated for single participant. | -8.600 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Calcium:Week 56, n=1,1,1,0 | -7.140 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -15.050 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Calcium:Week 60, n=1,1,1,0 | -5.100 (NA) — Standard deviation could not be calculated for single participant. | -1.060 (NA) — Standard deviation could not be calculated for single participant. | -11.830 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Calcium:Week 64, n=1,1,1,0 | -5.100 (NA) — Standard deviation could not be calculated for single participant. | 1.060 (NA) — Standard deviation could not be calculated for single participant. | -10.750 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Calcium:Week 68, n=1,0,1,0 | -2.040 (NA) — Standard deviation could not be calculated for single participant. |  | -8.600 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Calcium:Week 72, n=0,0,1,0 |  |  | -7.530 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Calcium:Week 76, n=0,0,1,0 |  |  | -11.830 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Calcium:Week 80, n=0,0,1,0 |  |  | -10.750 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Calcium:Week 84, n=0,0,1,0 |  |  | -6.450 (NA) — Standard deviation could not be calculated for single participant. |
  Calcium:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Calcium:Week 88, n=0,0,1,0 |  |  | -11.830 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  CO2:Week 1, n=0,0,3,1 |  |  | -4.130 (7.0589) | -4.170 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 2, n=11,11,12,2 | -7.175 (5.9450) | -1.014 (9.8790) | 0.698 (4.2233) | -8.330 (17.6777)
  CO2:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  CO2:Week 3, n=10,11,12,2 | -5.396 (8.3219) | -0.359 (9.4162) | 3.494 (8.5276) | 4.165 (11.7875)
  CO2:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  CO2:Week 4, n=10,11,11,2 | -4.261 (6.6572) | -0.885 (8.7334) | 1.185 (6.3365) | 6.250 (2.9416)
  CO2:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  CO2:Week 5, n=10,11,10,1 | -6.484 (6.1629) | -0.911 (13.3754) | -1.661 (7.0570) | 8.330 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 8, n=9,10,9,0: number analyzed (Participants) | 9 | 10 | 9 | 0
  CO2:Week 8, n=9,10,9,0 | -6.336 (7.2636) | 2.039 (9.9294) | 2.270 (6.9135) |
  CO2:Week 12, n=6,10,7,0: number analyzed (Participants) | 6 | 10 | 7 | 0
  CO2:Week 12, n=6,10,7,0 | -4.483 (11.0452) | 0.176 (8.2049) | -1.396 (7.6354) |
  CO2:Week 16, n=8,8,4,0: number analyzed (Participants) | 8 | 8 | 4 | 0
  CO2:Week 16, n=8,8,4,0 | -3.400 (5.6016) | -0.616 (11.9261) | -5.348 (3.8920) |
  CO2:Week 20, n=5,6,4,0: number analyzed (Participants) | 5 | 6 | 4 | 0
  CO2:Week 20, n=5,6,4,0 | -1.334 (2.9829) | 2.323 (11.0928) | 0.200 (4.9861) |
  CO2:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  CO2:Week 24, n=5,5,3,1 | -2.548 (8.4654) | -0.350 (10.9158) | -2.617 (2.2673) | 4.170 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  CO2:Week 28, n=5,4,3,1 | 0.454 (8.9936) | 1.625 (9.1644) | 0.050 (3.9252) | 8.330 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  CO2:Week 32, n=4,3,3,1 | -3.868 (9.1162) | -3.570 (3.5700) | 6.513 (5.9119) | 12.500 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  CO2:Week 36, n=3,1,3,1 | 0.277 (19.0084) | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 1.230 (5.9413) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  CO2:Week 40, n=1,2,2,1 | 3.330 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (5.0487) | 9.000 (1.4142) | -4.170 (NA) — Standard deviation could not be calculated for single participant.
  CO2:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  CO2:Week 44, n=1,2,2,0 | -6.670 (NA) — Standard deviation could not be calculated for single participant. | 3.570 (5.0487) | 2.000 (2.8284) |
  CO2:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  CO2:Week 48, n=1,1,1,0 | -3.330 (NA) — Standard deviation could not be calculated for single participant. | -3.570 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  CO2:Week 52, n=1,1,1,0 | 6.670 (NA) — Standard deviation could not be calculated for single participant. | 3.570 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  CO2:Week 56, n=1,1,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 14.290 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  CO2:Week 60, n=1,1,1,0 | -13.330 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  CO2:Week 64, n=1,1,1,0 | -6.670 (NA) — Standard deviation could not be calculated for single participant. | -10.710 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  CO2:Week 68, n=1,0,1,0 | -3.330 (NA) — Standard deviation could not be calculated for single participant. |  | 15.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  CO2:Week 72, n=0,0,1,0 |  |  | 5.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  CO2:Week 76, n=0,0,1,0 |  |  | 5.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  CO2:Week 80, n=0,0,1,0 |  |  | 20.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  CO2:Week 84, n=0,0,1,0 |  |  | 15.000 (NA) — Standard deviation could not be calculated for single participant. |
  CO2:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  CO2:Week 88, n=0,0,1,0 |  |  | -10.000 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Chloride:Week 1, n=0,0,3,1 |  |  | 0.000 (1.9600) | 4.000 (NA) — Standard deviation could not be calculated for single participant.
  Chloride:Week 2, n=11,11,12,1: number analyzed (Participants) | 11 | 11 | 12 | 1
  Chloride:Week 2, n=11,11,12,1 | 1.285 (2.5760) | 1.720 (2.0330) | 0.278 (2.1853) | -1.000 (NA) — Standard deviation could not be calculated for single participant.
  Chloride:Week 3, n=10,11,12,1: number analyzed (Participants) | 10 | 11 | 12 | 1
  Chloride:Week 3, n=10,11,12,1 | 1.110 (3.1963) | 2.169 (1.5618) | 1.042 (1.6055) | 1.000 (NA) — Standard deviation could not be calculated for single participant.
  Chloride:Week 4, n=10,11,11,1: number analyzed (Participants) | 10 | 11 | 11 | 1
  Chloride:Week 4, n=10,11,11,1 | 1.786 (1.2600) | 1.259 (1.9801) | 0.270 (1.2350) | 2.000 (NA) — Standard deviation could not be calculated for single participant.
  Chloride:Week 5, n=10,11,10,0: number analyzed (Participants) | 10 | 11 | 10 | 0
  Chloride:Week 5, n=10,11,10,0 | 1.038 (3.8548) | 0.825 (2.3370) | -0.495 (2.5736) |
  Chloride:Week 8, n=9,10,10,0: number analyzed (Participants) | 9 | 10 | 10 | 0
  Chloride:Week 8, n=9,10,10,0 | 1.342 (1.8157) | 0.514 (2.3134) | -1.613 (2.5122) |
  Chloride:Week 12, n=5,10,7,0: number analyzed (Participants) | 5 | 10 | 7 | 0
  Chloride:Week 12, n=5,10,7,0 | 2.218 (2.8158) | 1.564 (2.1107) | -1.077 (1.4931) |
  Chloride:Week 16, n=8,8,4,0: number analyzed (Participants) | 8 | 8 | 4 | 0
  Chloride:Week 16, n=8,8,4,0 | 1.379 (2.5654) | 1.979 (1.6634) | -0.755 (2.3017) |
  Chloride:Week 20, n=5,6,4,0: number analyzed (Participants) | 5 | 6 | 4 | 0
  Chloride:Week 20, n=5,6,4,0 | 1.818 (3.2011) | 2.842 (2.1684) | 0.470 (1.2655) |
  Chloride:Week 24, n=5,5,3,0: number analyzed (Participants) | 5 | 5 | 3 | 0
  Chloride:Week 24, n=5,5,3,0 | 1.016 (2.5283) | 0.204 (2.6191) | -0.590 (1.9337) |
  Chloride:Week 28, n=5,4,3,0: number analyzed (Participants) | 5 | 4 | 3 | 0
  Chloride:Week 28, n=5,4,3,0 | 2.012 (1.2468) | 1.515 (1.3092) | 0.050 (1.6282) |
  Chloride:Week 32, n=4,3,3,0: number analyzed (Participants) | 4 | 3 | 3 | 0
  Chloride:Week 32, n=4,3,3,0 | 2.230 (0.4359) | 2.027 (2.0200) | -0.377 (1.9704) |
  Chloride:Week 36, n=3,1,3,0: number analyzed (Participants) | 3 | 1 | 3 | 0
  Chloride:Week 36, n=3,1,3,0 | 1.703 (1.5832) | 1.020 (NA) — Standard deviation could not be calculated for single participant. | 1.283 (2.0455) |
  Chloride:Week 40, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Chloride:Week 40, n=1,2,2,0 | 2.970 (NA) — Standard deviation could not be calculated for single participant. | -2.560 (6.4771) | -0.500 (0.7071) |
  Chloride:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Chloride:Week 44, n=1,2,2,0 | 1.980 (NA) — Standard deviation could not be calculated for single participant. | 1.525 (0.7283) | 0.460 (0.6505) |
  Chloride:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Chloride:Week 48, n=1,1,1,0 | 3.960 (NA) — Standard deviation could not be calculated for single participant. | 3.030 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Chloride:Week 52, n=1,1,1,0 | 0.990 (NA) — Standard deviation could not be calculated for single participant. | 3.030 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Chloride:Week 56, n=1,1,1,0 | 2.970 (NA) — Standard deviation could not be calculated for single participant. | -1.010 (NA) — Standard deviation could not be calculated for single participant. | 1.830 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Chloride:Week 60, n=1,1,1,0 | 5.940 (NA) — Standard deviation could not be calculated for single participant. | -1.010 (NA) — Standard deviation could not be calculated for single participant. | 0.920 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Chloride:Week 64, n=1,1,1,0 | 3.960 (NA) — Standard deviation could not be calculated for single participant. | 4.040 (NA) — Standard deviation could not be calculated for single participant. | -0.920 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Chloride:Week 68, n=1,0,1,0 | 4.950 (NA) — Standard deviation could not be calculated for single participant. |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Chloride:Week 72, n=0,0,1,0 |  |  | -0.920 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Chloride:Week 76, n=0,0,1,0 |  |  | 1.830 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Chloride:Week 80, n=0,0,1,0 |  |  | -0.920 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Chloride:Week 84, n=0,0,1,0 |  |  | -1.830 (NA) — Standard deviation could not be calculated for single participant. |
  Chloride:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Chloride:Week 88, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Creatinine:Week 1, n=0,0,3,1 |  |  | 2.337 (0.9935) | 12.820 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 2, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Creatinine:Week 2, n=10,11,12,2 | 13.449 (12.6365) | 2.836 (13.7885) | 28.843 (62.8444) | 184.385 (248.7248)
  Creatinine:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Creatinine:Week 3, n=10,11,12,2 | 3.530 (6.0391) | 3.155 (12.3738) | 12.522 (28.5284) | 10.465 (8.7752)
  Creatinine:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Creatinine:Week 4, n=10,11,11,2 | 5.263 (13.2032) | -0.156 (11.9252) | 11.198 (29.2772) | 6.955 (17.3595)
  Creatinine:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Creatinine:Week 5, n=10,11,10,1 | 10.460 (13.3237) | -0.302 (13.6521) | 7.088 (13.6665) | -8.510 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Creatinine:Week 8, n=9,10,10,1 | 4.977 (8.1992) | -4.440 (10.4367) | 4.750 (7.8635) | -15.960 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  Creatinine:Week 12, n=7,10,7,1 | 13.411 (24.2292) | -1.289 (11.0396) | 2.236 (6.1696) | -13.830 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Creatinine:Week 16, n=8,8,4,1 | 7.920 (16.3323) | -5.519 (12.7681) | 2.875 (5.2082) | -6.380 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Creatinine:Week 20, n=5,6,4,1 | 8.414 (5.0623) | -3.007 (13.8034) | 10.315 (5.7571) | -2.130 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Creatinine:Week 24, n=5,5,3,1 | 14.184 (9.4608) | -11.006 (15.9134) | 4.737 (4.2811) | -5.320 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Creatinine:Week 28, n=5,4,3,1 | 12.888 (6.5007) | -12.093 (14.6604) | 2.520 (8.4940) | -1.060 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Creatinine:Week 32, n=4,3,3,1 | 11.690 (5.1478) | -17.913 (11.8535) | 11.320 (14.2430) | -7.450 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Creatinine:Week 36, n=3,1,3,1 | 10.500 (5.7663) | -30.530 (NA) — Standard deviation could not be calculated for single participant. | -25.153 (53.5998) | -18.090 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Creatinine:Week 40, n=1,2,2,1 | 20.000 (NA) — Standard deviation could not be calculated for single participant. | -13.230 (27.4357) | -0.245 (2.0294) | -12.770 (NA) — Standard deviation could not be calculated for single participant.
  Creatinine:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Creatinine:Week 44, n=1,2,2,0 | -6.000 (NA) — Standard deviation could not be calculated for single participant. | -13.775 (17.7413) | 8.470 (4.8508) |
  Creatinine:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Creatinine:Week 48, n=1,1,1,0 | 6.000 (NA) — Standard deviation could not be calculated for single participant. | -12.960 (NA) — Standard deviation could not be calculated for single participant. | -10.080 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Creatinine:Week 52, n=1,1,1,0 | 7.000 (NA) — Standard deviation could not be calculated for single participant. | -1.230 (NA) — Standard deviation could not be calculated for single participant. | 1.680 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Creatinine:Week 56, n=1,1,1,0 | -1.000 (NA) — Standard deviation could not be calculated for single participant. | -7.410 (NA) — Standard deviation could not be calculated for single participant. | 9.240 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Creatinine:Week 60, n=1,1,1,0 | 15.000 (NA) — Standard deviation could not be calculated for single participant. | -8.020 (NA) — Standard deviation could not be calculated for single participant. | 7.560 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Creatinine:Week 64, n=1,1,1,0 | 5.000 (NA) — Standard deviation could not be calculated for single participant. | 29.630 (NA) — Standard deviation could not be calculated for single participant. | -2.520 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Creatinine:Week 68, n=1,0,1,0 | -2.000 (NA) — Standard deviation could not be calculated for single participant. |  | -0.840 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine:Week 72, n=0,0,1,0 |  |  | 0.840 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine:Week 76, n=0,0,1,0 |  |  | -8.400 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine:Week 80, n=0,0,1,0 |  |  | -0.840 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine:Week 84, n=0,0,1,0 |  |  | -0.840 (NA) — Standard deviation could not be calculated for single participant. |
  Creatinine:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Creatinine:Week 88, n=0,0,1,0 |  |  | -13.450 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 1, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 1, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 2, n=4,4,6,1: number analyzed (Participants) | 4 | 4 | 6 | 1
  Direct bilirubin:Week 2, n=4,4,6,1 | 6.250 (65.7489) | -11.668 (23.3350) | -16.538 (40.5105) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Direct bilirubin:Week 3, n=3,2,6,1: number analyzed (Participants) | 3 | 2 | 6 | 1
  Direct bilirubin:Week 3, n=3,2,6,1 | -16.667 (28.8675) | 0.000 (0.0000) | -16.538 (40.5105) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Direct bilirubin:Week 4, n=3,6,6,1: number analyzed (Participants) | 3 | 6 | 6 | 1
  Direct bilirubin:Week 4, n=3,6,6,1 | -16.667 (28.8675) | 3.333 (32.0416) | 0.128 (63.0024) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Direct bilirubin:Week 5, n=3,6,5,0: number analyzed (Participants) | 3 | 6 | 5 | 0
  Direct bilirubin:Week 5, n=3,6,5,0 | -33.333 (28.8675) | -8.888 (14.4005) | -19.846 (44.3770) |
  Direct bilirubin:Week 8, n=3,5,4,0: number analyzed (Participants) | 3 | 5 | 4 | 0
  Direct bilirubin:Week 8, n=3,5,4,0 | -33.333 (38.1881) | 76.000 (133.7161) | 25.000 (50.0000) |
  Direct bilirubin:Week 12, n=1,5,3,0: number analyzed (Participants) | 1 | 5 | 3 | 0
  Direct bilirubin:Week 12, n=1,5,3,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 60.000 (134.1641) | 0.257 (99.6152) |
  Direct bilirubin:Week 16, n=2,4,2,0: number analyzed (Participants) | 2 | 4 | 2 | 0
  Direct bilirubin:Week 16, n=2,4,2,0 | -50.000 (35.3553) | 20.000 (54.1603) | -49.615 (70.1662) |
  Direct bilirubin:Week 20, n=0,2,1,0: number analyzed (Participants) | 0 | 2 | 1 | 0
  Direct bilirubin:Week 20, n=0,2,1,0 |  | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 24, n=0,3,1,0: number analyzed (Participants) | 0 | 3 | 1 | 0
  Direct bilirubin:Week 24, n=0,3,1,0 |  | -13.333 (23.0940) | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 28, n=0,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 0
  Direct bilirubin:Week 28, n=0,1,1,0 |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 32, n=0,2,1,0: number analyzed (Participants) | 0 | 2 | 1 | 0
  Direct bilirubin:Week 32, n=0,2,1,0 |  | -10.000 (14.1421) | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 36, n=0,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 0
  Direct bilirubin:Week 36, n=0,1,1,0 |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 40, n=0,2,0,0: number analyzed (Participants) | 0 | 2 | 0 | 0
  Direct bilirubin:Week 40, n=0,2,0,0 |  | -10.000 (14.1421) |  |
  Direct bilirubin:Week 44, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Direct bilirubin:Week 44, n=0,1,0,0 |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Direct bilirubin:Week 48, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Direct bilirubin:Week 48, n=0,1,0,0 |  | -20.000 (NA) — Standard deviation could not be calculated for single participant. |  |
  Direct bilirubin:Week 52, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Direct bilirubin:Week 56, n=0,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 0
  Direct bilirubin:Week 56, n=0,1,1,0 |  | -80.000 (NA) — Standard deviation could not be calculated for single participant. | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 60, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 60, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 64, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 64, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 68, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 68, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 72, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Direct bilirubin:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 76, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 80, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 84, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Direct bilirubin:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Direct bilirubin:Week 88, n=0,0,1,0 |  |  | -99.230 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 1, n=0,0,2,1: number analyzed (Participants) | 0 | 0 | 2 | 1
  Glucose:Week 1, n=0,0,2,1 |  |  | 25.745 (36.4089) | 40.630 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 2, n=11,10,12,2: number analyzed (Participants) | 11 | 10 | 12 | 2
  Glucose:Week 2, n=11,10,12,2 | -11.921 (14.9844) | 1.494 (21.6112) | -0.500 (13.1110) | 8.005 (4.8861)
  Glucose:Week 3, n=10,10,11,2: number analyzed (Participants) | 10 | 10 | 11 | 2
  Glucose:Week 3, n=10,10,11,2 | -4.956 (15.0667) | 1.229 (19.6823) | 2.856 (23.3024) | 35.985 (3.7547)
  Glucose:Week 4, n=9,10,10,2: number analyzed (Participants) | 9 | 10 | 10 | 2
  Glucose:Week 4, n=9,10,10,2 | -5.273 (9.5191) | 4.053 (31.5693) | -0.019 (11.9348) | 17.190 (11.0450)
  Glucose:Week 5, n=9,11,9,0: number analyzed (Participants) | 9 | 11 | 9 | 0
  Glucose:Week 5, n=9,11,9,0 | -2.012 (6.5775) | -2.482 (15.7553) | 1.737 (11.7985) |
  Glucose:Week 8, n=9,10,9,0: number analyzed (Participants) | 9 | 10 | 9 | 0
  Glucose:Week 8, n=9,10,9,0 | -5.971 (8.3770) | -4.807 (11.4303) | -2.250 (8.1208) |
  Glucose:Week 12, n=6,10,7,1: number analyzed (Participants) | 6 | 10 | 7 | 1
  Glucose:Week 12, n=6,10,7,1 | -4.812 (6.3454) | -3.481 (19.7216) | 2.353 (6.2058) | 18.180 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Glucose:Week 16, n=8,8,4,1 | -2.948 (8.0302) | -5.276 (10.6100) | 2.220 (10.1362) | 15.910 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Glucose:Week 20, n=5,6,4,1 | 2.184 (7.8557) | 0.290 (29.4058) | -4.715 (17.9623) | 13.640 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Glucose:Week 24, n=5,5,3,1 | -4.902 (14.4657) | 3.640 (22.3870) | 3.997 (9.6952) | 9.090 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Glucose:Week 28, n=5,4,3,1 | -0.288 (12.2744) | 11.950 (23.9058) | 3.610 (8.7790) | 9.090 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Glucose:Week 32, n=4,3,3,1 | 3.148 (21.6666) | -13.227 (15.6650) | 0.363 (2.7655) | 2.270 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Glucose:Week 36, n=3,1,3,1 | 0.247 (4.2508) | 20.620 (NA) — Standard deviation could not be calculated for single participant. | 3.320 (9.2103) | 13.640 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 40, n=1,1,2,1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Glucose:Week 40, n=1,1,2,1 | 18.180 (NA) — Standard deviation could not be calculated for single participant. | -10.310 (NA) — Standard deviation could not be calculated for single participant. | 3.485 (8.9308) | 22.730 (NA) — Standard deviation could not be calculated for single participant.
  Glucose:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Glucose:Week 44, n=1,2,2,0 | 17.170 (NA) — Standard deviation could not be calculated for single participant. | -7.955 (6.2438) | 3.485 (8.9308) |
  Glucose:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Glucose:Week 48, n=1,1,1,0 | 13.130 (NA) — Standard deviation could not be calculated for single participant. | -10.620 (NA) — Standard deviation could not be calculated for single participant. | -2.830 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Glucose:Week 52, n=1,1,1,0 | 7.070 (NA) — Standard deviation could not be calculated for single participant. | -3.540 (NA) — Standard deviation could not be calculated for single participant. | 2.830 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Glucose:Week 56, n=1,1,1,0 | -6.060 (NA) — Standard deviation could not be calculated for single participant. | 4.420 (NA) — Standard deviation could not be calculated for single participant. | 5.660 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Glucose:Week 60, n=1,1,1,0 | 2.020 (NA) — Standard deviation could not be calculated for single participant. | -15.930 (NA) — Standard deviation could not be calculated for single participant. | -1.890 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Glucose:Week 64, n=1,1,1,0 | -3.030 (NA) — Standard deviation could not be calculated for single participant. | 15.040 (NA) — Standard deviation could not be calculated for single participant. | -2.830 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Glucose:Week 68, n=1,0,1,0 | 10.100 (NA) — Standard deviation could not be calculated for single participant. |  | -0.940 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Glucose:Week 72, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Glucose:Week 76, n=0,0,1,0 |  |  | 9.430 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Glucose:Week 80, n=0,0,1,0 |  |  | -2.830 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Glucose:Week 84, n=0,0,1,0 |  |  | -2.830 (NA) — Standard deviation could not be calculated for single participant. |
  Glucose:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Glucose:Week 88, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Lactate dehydrogenase:Week 1, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 2, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 3, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 4, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 5, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 8, n=3,8,3,0: number analyzed (Participants) | 3 | 8 | 3 | 0
  Lactate dehydrogenase:Week 8, n=3,8,3,0 | 16.287 (3.9830) | 46.694 (62.1149) | 21.137 (14.3265) |
  Lactate dehydrogenase:Week 12, n=2,8,4,0: number analyzed (Participants) | 2 | 8 | 4 | 0
  Lactate dehydrogenase:Week 12, n=2,8,4,0 | 12.870 (3.0123) | 39.709 (54.5987) | 31.353 (17.3375) |
  Lactate dehydrogenase:Week 16, n=2,6,3,1: number analyzed (Participants) | 2 | 6 | 3 | 1
  Lactate dehydrogenase:Week 16, n=2,6,3,1 | 14.965 (10.5571) | 53.818 (83.5554) | 37.677 (22.5797) | 36.870 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 20, n=2,5,3,1: number analyzed (Participants) | 2 | 5 | 3 | 1
  Lactate dehydrogenase:Week 20, n=2,5,3,1 | 13.145 (7.9832) | 7.232 (21.7161) | 35.440 (24.8959) | 14.290 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 24, n=2,4,2,1: number analyzed (Participants) | 2 | 4 | 2 | 1
  Lactate dehydrogenase:Week 24, n=2,4,2,1 | 13.415 (5.7064) | 81.540 (74.2387) | 22.745 (2.9486) | 20.280 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 28, n=2,3,1,1: number analyzed (Participants) | 2 | 3 | 1 | 1
  Lactate dehydrogenase:Week 28, n=2,3,1,1 | 10.485 (5.0982) | 24.857 (27.3567) | 26.850 (NA) — Standard deviation could not be calculated for single participant. | 18.890 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 32, n=2,3,1,1: number analyzed (Participants) | 2 | 3 | 1 | 1
  Lactate dehydrogenase:Week 32, n=2,3,1,1 | 14.000 (16.2635) | 63.040 (60.6775) | 13.150 (NA) — Standard deviation could not be calculated for single participant. | 33.180 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 36, n=2,1,0,1: number analyzed (Participants) | 2 | 1 | 0 | 1
  Lactate dehydrogenase:Week 36, n=2,1,0,1 | 20.795 (16.1432) | 38.670 (NA) — Standard deviation could not be calculated for single participant. |  | 12.440 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 40, n=0,2,0,1: number analyzed (Participants) | 0 | 2 | 0 | 1
  Lactate dehydrogenase:Week 40, n=0,2,0,1 |  | 75.840 (84.5983) |  | 11.980 (NA) — Standard deviation could not be calculated for single participant.
  Lactate dehydrogenase:Week 44, n=0,2,0,0: number analyzed (Participants) | 0 | 2 | 0 | 0
  Lactate dehydrogenase:Week 44, n=0,2,0,0 |  | 31.175 (79.3586) |  |
  Lactate dehydrogenase:Week 48, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Lactate dehydrogenase:Week 48, n=0,1,0,0 |  | 80.800 (NA) — Standard deviation could not be calculated for single participant. |  |
  Lactate dehydrogenase:Week 52, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Lactate dehydrogenase:Week 52, n=0,1,0,0 |  | -42.640 (NA) — Standard deviation could not be calculated for single participant. |  |
  Lactate dehydrogenase:Week 56, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Lactate dehydrogenase:Week 56, n=0,1,0,0 |  | -44.390 (NA) — Standard deviation could not be calculated for single participant. |  |
  Lactate dehydrogenase:Week 60, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Lactate dehydrogenase:Week 60, n=0,1,0,0 |  | -41.900 (NA) — Standard deviation could not be calculated for single participant. |  |
  Lactate dehydrogenase:Week 64, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Lactate dehydrogenase:Week 64, n=0,1,0,0 |  | -49.130 (NA) — Standard deviation could not be calculated for single participant. |  |
  Lactate dehydrogenase:Week 68, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 72, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 76, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 80, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 84, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Lactate dehydrogenase:Week 88, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Magnesium:Week 1, n=0,0,3,0: number analyzed (Participants) | 0 | 0 | 3 | 0
  Magnesium:Week 1, n=0,0,3,0 |  |  | -2.013 (10.2561) |
  Magnesium:Week 2, n=9,10,11,2: number analyzed (Participants) | 9 | 10 | 11 | 2
  Magnesium:Week 2, n=9,10,11,2 | 3.687 (10.9267) | 4.413 (5.0742) | 3.593 (13.9856) | -3.205 (10.3591)
  Magnesium:Week 3, n=8,11,11,2: number analyzed (Participants) | 8 | 11 | 11 | 2
  Magnesium:Week 3, n=8,11,11,2 | -1.633 (4.7088) | 6.602 (10.8819) | -1.808 (12.3971) | -24.200 (32.7673)
  Magnesium:Week 4, n=8,11,10,2: number analyzed (Participants) | 8 | 11 | 10 | 2
  Magnesium:Week 4, n=8,11,10,2 | 4.104 (5.7486) | 4.971 (7.7656) | 1.254 (8.2818) | -20.430 (15.7685)
  Magnesium:Week 5, n=10,11,9,1: number analyzed (Participants) | 10 | 11 | 9 | 1
  Magnesium:Week 5, n=10,11,9,1 | -1.521 (6.3803) | 5.014 (12.0008) | 5.071 (8.7326) | -7.220 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 8, n=8,10,9,0: number analyzed (Participants) | 8 | 10 | 9 | 0
  Magnesium:Week 8, n=8,10,9,0 | -0.370 (5.3051) | 3.458 (6.0669) | 3.469 (7.9381) |
  Magnesium:Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  Magnesium:Week 12, n=7,10,7,1 | 0.904 (3.4827) | 1.288 (10.5039) | -1.844 (7.2017) | -3.090 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Magnesium:Week 16, n=8,8,4,1 | 4.311 (5.1089) | 0.045 (10.0780) | -3.303 (9.9862) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Magnesium:Week 20, n=5,6,4,1 | -2.720 (6.2671) | 3.043 (6.1070) | -5.430 (4.0591) | -2.060 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Magnesium:Week 24, n=5,5,3,1 | -1.790 (6.7929) | 1.390 (11.0108) | -5.453 (1.6991) | -5.150 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 28, n=5,3,3,1: number analyzed (Participants) | 5 | 3 | 3 | 1
  Magnesium:Week 28, n=5,3,3,1 | -0.512 (3.6523) | 9.137 (12.3852) | -5.433 (7.6708) | -9.280 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Magnesium:Week 32, n=4,3,3,1 | -0.303 (3.0947) | 9.400 (15.8067) | -2.843 (4.5798) | 1.030 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Magnesium:Week 36, n=3,1,3,1 | -2.917 (5.0518) | 13.330 (NA) — Standard deviation could not be calculated for single participant. | 1.673 (3.8829) | -3.090 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 40, n=1,1,2,1: number analyzed (Participants) | 1 | 1 | 2 | 1
  Magnesium:Week 40, n=1,1,2,1 | 10.000 (NA) — Standard deviation could not be calculated for single participant. | 13.330 (NA) — Standard deviation could not be calculated for single participant. | -2.780 (3.9315) | -3.090 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Magnesium:Week 44, n=1,2,2,0 | -5.000 (NA) — Standard deviation could not be calculated for single participant. | 2.315 (15.5776) | 0.000 (0.0000) |
  Magnesium:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Magnesium:Week 48, n=1,1,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -4.350 (NA) — Standard deviation could not be calculated for single participant. | -13.040 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Magnesium:Week 52, n=1,1,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -8.700 (NA) — Standard deviation could not be calculated for single participant. | -13.040 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Magnesium:Week 56, n=1,1,1,0 | -5.000 (NA) — Standard deviation could not be calculated for single participant. | -8.700 (NA) — Standard deviation could not be calculated for single participant. | 8.700 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Magnesium:Week 60, n=1,1,1,0 | -5.000 (NA) — Standard deviation could not be calculated for single participant. | 4.350 (NA) — Standard deviation could not be calculated for single participant. | -4.350 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Magnesium:Week 64, n=1,1,1,0 | 5.000 (NA) — Standard deviation could not be calculated for single participant. | -4.350 (NA) — Standard deviation could not be calculated for single participant. | -4.350 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Magnesium:Week 68, n=1,0,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium:Week 72, n=0,0,1,0 |  |  | -4.350 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium:Week 76, n=0,0,1,0 |  |  | -8.700 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium:Week 80, n=0,0,1,0 |  |  | -4.350 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium:Week 84, n=0,0,1,0 |  |  | -4.350 (NA) — Standard deviation could not be calculated for single participant. |
  Magnesium:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Magnesium:Week 88, n=0,0,1,0 |  |  | -17.390 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Potassium:Week 1, n=0,0,3,1 |  |  | 2.560 (4.7011) | 10.870 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 2, n=11,11,12,2 | 6.295 (11.2391) | 0.394 (10.9402) | -2.844 (9.6594) | -1.085 (13.8381)
  Potassium:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Potassium:Week 3, n=10,11,12,2 | 4.095 (9.1369) | -0.879 (5.4861) | 0.837 (7.9003) | -10.870 (6.1518)
  Potassium:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Potassium:Week 4, n=10,11,11,2 | 5.295 (12.9147) | 2.234 (10.6975) | -2.279 (8.2128) | -1.085 (1.5344)
  Potassium:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Potassium:Week 5, n=10,11,10,1 | 0.613 (13.4203) | 3.677 (8.4593) | 0.479 (6.7468) | -4.350 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Potassium:Week 8, n=9,10,10,1 | 3.551 (10.1989) | -0.714 (10.4143) | -2.574 (8.8434) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 12, n=6,10,7,1: number analyzed (Participants) | 6 | 10 | 7 | 1
  Potassium:Week 12, n=6,10,7,1 | 6.910 (7.7994) | 0.801 (9.1329) | 0.097 (6.5124) | -4.350 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Potassium:Week 16, n=8,8,4,1 | 3.099 (11.1450) | 0.391 (7.4310) | 0.825 (7.0552) | 4.350 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Potassium:Week 20, n=5,6,4,1 | 7.054 (6.5355) | -1.055 (8.0880) | 3.608 (7.3186) | -2.170 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Potassium:Week 24, n=5,5,3,1 | 4.250 (15.2421) | -2.684 (11.5575) | 2.383 (2.4420) | -4.350 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Potassium:Week 28, n=5,4,3,1 | 4.134 (13.7038) | -1.040 (11.5877) | 1.793 (7.5585) | -4.350 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Potassium:Week 32, n=4,3,3,1 | 10.555 (11.6304) | 2.973 (14.6875) | -3.143 (2.7272) | 4.350 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Potassium:Week 36, n=3,1,3,1 | 5.650 (12.0712) | 18.920 (NA) — Standard deviation could not be calculated for single participant. | 3.253 (5.6349) | -6.520 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Potassium:Week 40, n=1,2,2,1 | 17.070 (NA) — Standard deviation could not be calculated for single participant. | 0.265 (7.2761) | -2.440 (3.4507) | -8.700 (NA) — Standard deviation could not be calculated for single participant.
  Potassium:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Potassium:Week 44, n=1,2,2,0 | 12.200 (NA) — Standard deviation could not be calculated for single participant. | 10.550 (8.0186) | 5.935 (1.9587) |
  Potassium:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Potassium:Week 48, n=1,1,1,0 | 24.390 (NA) — Standard deviation could not be calculated for single participant. | -4.880 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Potassium:Week 52, n=1,1,1,0 | 24.390 (NA) — Standard deviation could not be calculated for single participant. | -2.440 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Potassium:Week 56, n=1,1,1,0 | -2.440 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -2.270 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Potassium:Week 60, n=1,1,1,0 | 12.200 (NA) — Standard deviation could not be calculated for single participant. | -2.440 (NA) — Standard deviation could not be calculated for single participant. | -4.550 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Potassium:Week 64, n=1,1,1,0 | 24.390 (NA) — Standard deviation could not be calculated for single participant. | -12.200 (NA) — Standard deviation could not be calculated for single participant. | -4.550 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Potassium:Week 68, n=1,0,1,0 | 29.270 (NA) — Standard deviation could not be calculated for single participant. |  | 2.270 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium:Week 72, n=0,0,1,0 |  |  | -2.270 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium:Week 76, n=0,0,1,0 |  |  | -4.550 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium:Week 80, n=0,0,1,0 |  |  | 4.550 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium:Week 84, n=0,0,1,0 |  |  | -2.270 (NA) — Standard deviation could not be calculated for single participant. |
  Potassium:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Potassium:Week 88, n=0,0,1,0 |  |  | -6.820 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Sodium:Week 1, n=0,0,3,1 |  |  | -1.657 (2.2823) | 2.860 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 2, n=11,11,12,2 | 0.013 (1.8096) | -0.370 (1.9173) | 0.266 (1.7336) | 0.000 (2.0223)
  Sodium:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Sodium:Week 3, n=10,11,12,2 | 0.311 (1.8340) | 0.009 (1.5263) | 0.308 (1.6247) | 1.430 (2.0223)
  Sodium:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Sodium:Week 4, n=10,11,11,2 | 0.383 (1.4528) | -0.178 (1.9638) | 0.545 (1.5916) | 0.710 (0.0000)
  Sodium:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Sodium:Week 5, n=10,11,10,1 | 0.890 (1.2598) | -0.255 (1.2916) | -0.791 (1.5272) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Sodium:Week 8, n=9,10,10,1 | 0.312 (1.9462) | -0.132 (1.5679) | -0.643 (1.5180) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 12, n=6,10,7,1: number analyzed (Participants) | 6 | 10 | 7 | 1
  Sodium:Week 12, n=6,10,7,1 | 0.597 (1.2596) | 0.080 (1.3734) | -0.816 (1.0457) | 2.140 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Sodium:Week 16, n=8,8,4,1 | 0.643 (1.4831) | 0.009 (1.3395) | -1.773 (2.7477) | 2.140 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Sodium:Week 20, n=5,6,4,1 | 1.904 (1.3431) | 0.722 (0.6509) | -0.173 (1.2213) | -0.710 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Sodium:Week 24, n=5,5,3,1 | 0.584 (1.4250) | -0.424 (1.5620) | -0.953 (0.4215) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Sodium:Week 28, n=5,4,3,1 | 1.606 (0.9562) | -0.538 (0.3584) | -0.237 (1.4852) | -0.710 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Sodium:Week 32, n=4,3,3,1 | 0.363 (0.9515) | 0.953 (1.8133) | -0.233 (1.4932) | -0.710 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Sodium:Week 36, n=3,1,3,1 | 0.737 (1.4550) | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -0.237 (0.4099) | 2.140 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Sodium:Week 40, n=1,2,2,1 | 2.960 (NA) — Standard deviation could not be calculated for single participant. | -1.385 (5.0134) | -1.070 (1.5132) | 1.430 (NA) — Standard deviation could not be calculated for single participant.
  Sodium:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Sodium:Week 44, n=1,2,2,0 | 2.220 (NA) — Standard deviation could not be calculated for single participant. | 0.350 (0.4950) | 0.725 (2.0294) |
  Sodium:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Sodium:Week 48, n=1,1,1,0 | 2.220 (NA) — Standard deviation could not be calculated for single participant. | 4.320 (NA) — Standard deviation could not be calculated for single participant. | -1.440 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Sodium:Week 52, n=1,1,1,0 | 2.220 (NA) — Standard deviation could not be calculated for single participant. | 0.720 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Sodium:Week 56, n=1,1,1,0 | 3.700 (NA) — Standard deviation could not be calculated for single participant. | -1.440 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Sodium:Week 60, n=1,1,1,0 | 2.220 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Sodium:Week 64, n=1,1,1,0 | 2.220 (NA) — Standard deviation could not be calculated for single participant. | 0.720 (NA) — Standard deviation could not be calculated for single participant. | -2.160 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Sodium:Week 68, n=1,0,1,0 | 3.700 (NA) — Standard deviation could not be calculated for single participant. |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Sodium:Week 72, n=0,0,1,0 |  |  | -0.720 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Sodium:Week 76, n=0,0,1,0 |  |  | 0.720 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Sodium:Week 80, n=0,0,1,0 |  |  | 0.720 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Sodium:Week 84, n=0,0,1,0 |  |  | -0.720 (NA) — Standard deviation could not be calculated for single participant. |
  Sodium:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Sodium:Week 88, n=0,0,1,0 |  |  | -0.720 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Total bilirubin:Week 1, n=0,0,3,1 |  |  | -42.590 (8.4876) | -50.000 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 2, n=11,11,12,2 | -14.740 (19.0474) | -12.683 (35.0603) | -0.972 (48.2811) | -47.220 (3.9315)
  Total bilirubin:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Total bilirubin:Week 3, n=10,11,12,2 | -14.679 (18.3507) | -1.768 (31.6024) | -10.532 (29.0132) | -6.945 (25.5336)
  Total bilirubin:Week 4, n=10,11,11,2: number analyzed (Participants) | 10 | 11 | 11 | 2
  Total bilirubin:Week 4, n=10,11,11,2 | -2.488 (26.5820) | 24.492 (57.3828) | 2.855 (25.9280) | 12.500 (17.6777)
  Total bilirubin:Week 5, n=10,11,10,1: number analyzed (Participants) | 10 | 11 | 10 | 1
  Total bilirubin:Week 5, n=10,11,10,1 | -0.500 (19.7836) | 12.879 (40.0010) | 13.944 (48.2067) | -22.220 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 8, n=9,10,10,1: number analyzed (Participants) | 9 | 10 | 10 | 1
  Total bilirubin:Week 8, n=9,10,10,1 | -3.744 (22.8000) | 45.680 (62.1644) | 21.972 (40.2576) | -55.560 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  Total bilirubin:Week 12, n=7,10,7,1 | -6.276 (27.3764) | 20.223 (39.6273) | 4.364 (18.2751) | -44.440 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Total bilirubin:Week 16, n=8,8,4,1 | -5.739 (13.8572) | 16.473 (48.6051) | -4.165 (20.9713) | -44.440 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 20, n=5,6,4,1: number analyzed (Participants) | 5 | 6 | 4 | 1
  Total bilirubin:Week 20, n=5,6,4,1 | 4.454 (23.8194) | -15.500 (23.5242) | -15.973 (11.1972) | -22.220 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Total bilirubin:Week 24, n=5,5,3,1 | -14.500 (8.7321) | -0.714 (56.6292) | -19.443 (17.3459) | -11.110 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Total bilirubin:Week 28, n=5,4,3,1 | -3.182 (22.6771) | -4.165 (20.9713) | 0.000 (0.0000) | -22.220 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Total bilirubin:Week 32, n=4,3,3,1 | -12.215 (23.6747) | -13.890 (12.7297) | 1.853 (13.9824) | -33.330 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Total bilirubin:Week 36, n=3,1,3,1 | 9.167 (18.7639) | 50.000 (NA) — Standard deviation could not be calculated for single participant. | -12.963 (11.5645) | -44.440 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Total bilirubin:Week 40, n=1,2,2,1 | -37.500 (NA) — Standard deviation could not be calculated for single participant. | -16.665 (23.5679) | -25.000 (35.3553) | -55.560 (NA) — Standard deviation could not be calculated for single participant.
  Total bilirubin:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Total bilirubin:Week 44, n=1,2,2,0 | -25.000 (NA) — Standard deviation could not be calculated for single participant. | 8.335 (58.9232) | -18.055 (9.8217) |
  Total bilirubin:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total bilirubin:Week 48, n=1,1,1,0 | -25.000 (NA) — Standard deviation could not be calculated for single participant. | -16.670 (NA) — Standard deviation could not be calculated for single participant. | -50.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total bilirubin:Week 52, n=1,1,1,0 | -12.500 (NA) — Standard deviation could not be calculated for single participant. | -50.000 (NA) — Standard deviation could not be calculated for single participant. | -50.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total bilirubin:Week 56, n=1,1,1,0 | -50.000 (NA) — Standard deviation could not be calculated for single participant. | -33.330 (NA) — Standard deviation could not be calculated for single participant. | -25.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total bilirubin:Week 60, n=1,1,1,0 | -37.500 (NA) — Standard deviation could not be calculated for single participant. | -66.670 (NA) — Standard deviation could not be calculated for single participant. | -25.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total bilirubin:Week 64, n=1,1,1,0 | -37.500 (NA) — Standard deviation could not be calculated for single participant. | -66.670 (NA) — Standard deviation could not be calculated for single participant. | -50.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Total bilirubin:Week 68, n=1,0,1,0 | -25.000 (NA) — Standard deviation could not be calculated for single participant. |  | -50.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total bilirubin:Week 72, n=0,0,1,0 |  |  | -25.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total bilirubin:Week 76, n=0,0,1,0 |  |  | -25.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total bilirubin:Week 80, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total bilirubin:Week 84, n=0,0,1,0 |  |  | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total bilirubin:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total bilirubin:Week 88, n=0,0,1,0 |  |  | 50.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  Total protein:Week 1, n=0,0,3,1 |  |  | 1.380 (2.8026) | 3.170 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 2, n=11,11,12,1: number analyzed (Participants) | 11 | 11 | 12 | 1
  Total protein:Week 2, n=11,11,12,1 | 2.140 (7.3161) | -14.885 (32.7433) | 82.059 (278.6333) | -1.590 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 3, n=10,11,12,2: number analyzed (Participants) | 10 | 11 | 12 | 2
  Total protein:Week 3, n=10,11,12,2 | -2.260 (5.4555) | -5.132 (18.9226) | 60.186 (206.7731) | -0.110 (2.0930)
  Total protein:Week 4, n=10,10,11,2: number analyzed (Participants) | 10 | 10 | 11 | 2
  Total protein:Week 4, n=10,10,11,2 | -0.132 (4.5645) | -5.886 (18.8830) | -0.086 (4.6004) | -9.090 (5.1053)
  Total protein:Week 5, n=9,11,10,0: number analyzed (Participants) | 9 | 11 | 10 | 0
  Total protein:Week 5, n=9,11,10,0 | -8.962 (26.1684) | -5.207 (16.4970) | 1.943 (6.8329) |
  Total protein:Week 8, n=8,10,10,0: number analyzed (Participants) | 8 | 10 | 10 | 0
  Total protein:Week 8, n=8,10,10,0 | 0.981 (3.3039) | -7.914 (16.5027) | 2.247 (6.1649) |
  Total protein:Week 12, n=7,10,7,1: number analyzed (Participants) | 7 | 10 | 7 | 1
  Total protein:Week 12, n=7,10,7,1 | 0.570 (5.5899) | -7.764 (17.4075) | 1.009 (4.6858) | -2.740 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Total protein:Week 16, n=8,8,4,1 | 0.336 (6.3130) | -10.768 (17.9309) | -4.268 (6.0907) | 5.480 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 20, n=5,6,3,1: number analyzed (Participants) | 5 | 6 | 3 | 1
  Total protein:Week 20, n=5,6,3,1 | -1.520 (7.6530) | -2.397 (4.8249) | 2.390 (3.3674) | 4.110 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Total protein:Week 24, n=5,5,3,1 | -0.368 (6.3631) | -1.748 (6.0092) | -3.713 (7.2790) | 2.740 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 28, n=5,4,3,1: number analyzed (Participants) | 5 | 4 | 3 | 1
  Total protein:Week 28, n=5,4,3,1 | 0.168 (5.4900) | -3.243 (3.2436) | 0.000 (6.2070) | 4.110 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Total protein:Week 32, n=4,3,3,1 | 0.490 (6.4817) | -4.220 (1.4543) | -1.160 (12.5647) | 2.740 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 36, n=2,1,3,1: number analyzed (Participants) | 2 | 1 | 3 | 1
  Total protein:Week 36, n=2,1,3,1 | -0.580 (2.9981) | -3.170 (NA) — Standard deviation could not be calculated for single participant. | 0.447 (4.3016) | 4.110 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Total protein:Week 40, n=1,2,2,1 | -4.050 (NA) — Standard deviation could not be calculated for single participant. | -7.935 (11.2218) | -7.115 (8.1247) | -2.740 (NA) — Standard deviation could not be calculated for single participant.
  Total protein:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  Total protein:Week 44, n=1,2,2,0 | -1.350 (NA) — Standard deviation could not be calculated for single participant. | -6.380 (2.2062) | -0.205 (13.8522) |
  Total protein:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total protein:Week 48, n=1,1,1,0 | -5.410 (NA) — Standard deviation could not be calculated for single participant. | -1.200 (NA) — Standard deviation could not be calculated for single participant. | -11.430 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total protein:Week 52, n=1,1,1,0 | -2.700 (NA) — Standard deviation could not be calculated for single participant. | -6.020 (NA) — Standard deviation could not be calculated for single participant. | -8.570 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total protein:Week 56, n=1,1,1,0 | -6.760 (NA) — Standard deviation could not be calculated for single participant. | -9.640 (NA) — Standard deviation could not be calculated for single participant. | -10.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total protein:Week 60, n=1,1,1,0 | -2.700 (NA) — Standard deviation could not be calculated for single participant. | -6.020 (NA) — Standard deviation could not be calculated for single participant. | -8.570 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Total protein:Week 64, n=1,1,1,0 | -6.760 (NA) — Standard deviation could not be calculated for single participant. | -9.640 (NA) — Standard deviation could not be calculated for single participant. | -8.570 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Total protein:Week 68, n=1,0,1,0 | -5.410 (NA) — Standard deviation could not be calculated for single participant. |  | -11.430 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total protein:Week 72, n=0,0,1,0 |  |  | -10.000 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total protein:Week 76, n=0,0,1,0 |  |  | -17.140 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total protein:Week 80, n=0,0,1,0 |  |  | -8.570 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total protein:Week 84, n=0,0,1,0 |  |  | -5.710 (NA) — Standard deviation could not be calculated for single participant. |
  Total protein:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Total protein:Week 88, n=0,0,1,0 |  |  | -11.430 (NA) — Standard deviation could not be calculated for single participant. |

7. Primary Outcome: Percent Change From Baseline in Chemistry Parameters During Combination Treatment Period: Blood Urea Nitrogen (BUN), Uric Acid
Description: Blood samples were collected to analyze the chemistry parameters: BUN and uric acid. Baseline value is the latest GSK2636771 pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100 multiplied by (post-Baseline visit value minus Baseline divided by Baseline).
Time Frame: Baseline (Day 1), Weeks 1, 2,3,4,5,8,12,16,20,24,28,32,36,40,44,48,52,56,60,64,68,72,76,80,84 and 88
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 10 | 11 | 12 | 2
Percent change
  BUN:Week 1, n=0,0,3,1: number analyzed (Participants) | 0 | 0 | 3 | 1
  BUN:Week 1, n=0,0,3,1 |  |  | -10.227 (9.3008) | 18.180 (NA) — Standard deviation could not be calculated for single participant.
  BUN:Week 2, n=10,11,12,1: number analyzed (Participants) | 10 | 11 | 12 | 1
  BUN:Week 2, n=10,11,12,1 | -5.741 (24.5046) | -7.622 (18.4784) | 1.848 (44.3336) | 236.360 (NA) — Standard deviation could not be calculated for single participant.
  BUN:Week 3, n=8,11,12,1: number analyzed (Participants) | 8 | 11 | 12 | 1
  BUN:Week 3, n=8,11,12,1 | -10.699 (18.9576) | -12.921 (8.9324) | -9.143 (22.4881) | 45.450 (NA) — Standard deviation could not be calculated for single participant.
  BUN:Week 4, n=9,11,11,1: number analyzed (Participants) | 9 | 11 | 11 | 1
  BUN:Week 4, n=9,11,11,1 | -12.330 (16.4809) | -13.030 (17.8055) | -11.637 (19.2345) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  BUN:Week 5, n=9,11,10,0: number analyzed (Participants) | 9 | 11 | 10 | 0
  BUN:Week 5, n=9,11,10,0 | -14.012 (12.6452) | -8.568 (18.3100) | 1.857 (19.8509) |
  BUN:Week 8, n=9,10,10,0: number analyzed (Participants) | 9 | 10 | 10 | 0
  BUN:Week 8, n=9,10,10,0 | -8.916 (22.6106) | -16.238 (16.8508) | -12.537 (14.8918) |
  BUN:Week 12, n=6,10,7,0: number analyzed (Participants) | 6 | 10 | 7 | 0
  BUN:Week 12, n=6,10,7,0 | 0.090 (20.4882) | -12.186 (20.8205) | -10.536 (18.6180) |
  BUN:Week 16, n=8,8,4,0: number analyzed (Participants) | 8 | 8 | 4 | 0
  BUN:Week 16, n=8,8,4,0 | -5.259 (14.6735) | -18.011 (12.0206) | -5.560 (22.5383) |
  BUN:Week 20, n=5,6,4,0: number analyzed (Participants) | 5 | 6 | 4 | 0
  BUN:Week 20, n=5,6,4,0 | -9.110 (12.9929) | -6.380 (21.2869) | -6.910 (20.6469) |
  BUN:Week 24, n=5,5,3,0: number analyzed (Participants) | 5 | 5 | 3 | 0
  BUN:Week 24, n=5,5,3,0 | -4.036 (9.0958) | -13.412 (29.3172) | 7.450 (8.7505) |
  BUN:Week 28, n=5,4,3,0: number analyzed (Participants) | 5 | 4 | 3 | 0
  BUN:Week 28, n=5,4,3,0 | -11.508 (10.1606) | -21.773 (9.5686) | 12.603 (15.4411) |
  BUN:Week 32, n=4,3,3,0: number analyzed (Participants) | 4 | 3 | 3 | 0
  BUN:Week 32, n=4,3,3,0 | -8.163 (11.5276) | -7.553 (30.6672) | -16.567 (12.1882) |
  BUN:Week 36, n=3,1,3,0: number analyzed (Participants) | 3 | 1 | 3 | 0
  BUN:Week 36, n=3,1,3,0 | -7.593 (12.0178) | 0.000 (NA) — Standard deviation could not be calculated for single participant. | 1.970 (29.1203) |
  BUN:Week 40, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  BUN:Week 40, n=1,2,2,0 | 16.670 (NA) — Standard deviation could not be calculated for single participant. | 27.885 (90.2056) | -7.275 (3.8537) |
  BUN:Week 44, n=1,2,2,0: number analyzed (Participants) | 1 | 2 | 2 | 0
  BUN:Week 44, n=1,2,2,0 | -5.560 (NA) — Standard deviation could not be calculated for single participant. | -26.285 (13.5977) | -6.060 (15.0048) |
  BUN:Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  BUN:Week 48, n=1,1,1,0 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -17.950 (NA) — Standard deviation could not be calculated for single participant. | -10.000 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 52, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  BUN:Week 52, n=1,1,1,0 | 5.560 (NA) — Standard deviation could not be calculated for single participant. | -23.080 (NA) — Standard deviation could not be calculated for single participant. | -3.330 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 56, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  BUN:Week 56, n=1,1,1,0 | -22.220 (NA) — Standard deviation could not be calculated for single participant. | -30.770 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 60, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  BUN:Week 60, n=1,1,1,0 | 55.560 (NA) — Standard deviation could not be calculated for single participant. | -7.690 (NA) — Standard deviation could not be calculated for single participant. | -23.330 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 64, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  BUN:Week 64, n=1,1,1,0 | 5.560 (NA) — Standard deviation could not be calculated for single participant. | -15.380 (NA) — Standard deviation could not be calculated for single participant. | -16.670 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  BUN:Week 68, n=1,0,1,0 | -11.110 (NA) — Standard deviation could not be calculated for single participant. |  | -26.670 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  BUN:Week 72, n=0,0,1,0 |  |  | -23.330 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  BUN:Week 76, n=0,0,1,0 |  |  | -20.000 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  BUN:Week 80, n=0,0,1,0 |  |  | -26.670 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  BUN:Week 84, n=0,0,1,0 |  |  | -10.000 (NA) — Standard deviation could not be calculated for single participant. |
  BUN:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  BUN:Week 88, n=0,0,1,0 |  |  | -70.000 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 1, n=0,0,3,0: number analyzed (Participants) | 0 | 0 | 3 | 0
  Uric acid:Week 1, n=0,0,3,0 |  |  | 6.513 (3.2031) |
  Uric acid:Week 2, n=8,10,11,2: number analyzed (Participants) | 8 | 10 | 11 | 2
  Uric acid:Week 2, n=8,10,11,2 | -11.656 (33.0629) | 158.135 (499.1483) | 13.357 (26.0799) | 71.090 (46.6549)
  Uric acid:Week 3, n=7,9,11,2: number analyzed (Participants) | 7 | 9 | 11 | 2
  Uric acid:Week 3, n=7,9,11,2 | -4.581 (14.8856) | 154.651 (480.5708) | 0.284 (14.9816) | 25.170 (38.4808)
  Uric acid:Week 4, n=7,11,10,1: number analyzed (Participants) | 7 | 11 | 10 | 1
  Uric acid:Week 4, n=7,11,10,1 | 1.053 (12.8059) | -3.509 (7.9426) | 4.436 (22.8767) | 14.290 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 5, n=9,11,9,0: number analyzed (Participants) | 9 | 11 | 9 | 0
  Uric acid:Week 5, n=9,11,9,0 | 1.676 (8.0283) | 139.415 (481.0482) | 0.532 (10.9365) |
  Uric acid:Week 8, n=8,10,9,0: number analyzed (Participants) | 8 | 10 | 9 | 0
  Uric acid:Week 8, n=8,10,9,0 | 3.543 (16.5957) | -7.224 (9.7223) | 0.440 (10.9092) |
  Uric acid:Week 12, n=6,10,6,1: number analyzed (Participants) | 6 | 10 | 6 | 1
  Uric acid:Week 12, n=6,10,6,1 | 4.578 (19.8500) | -1.403 (5.7519) | -0.210 (12.5985) | 28.570 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 16, n=8,8,4,1: number analyzed (Participants) | 8 | 8 | 4 | 1
  Uric acid:Week 16, n=8,8,4,1 | 3.146 (8.8330) | -7.384 (8.5001) | -3.473 (5.4805) | 52.380 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 20, n=5,5,4,1: number analyzed (Participants) | 5 | 5 | 4 | 1
  Uric acid:Week 20, n=5,5,4,1 | 2.232 (5.4135) | -1.796 (8.1659) | 1.920 (10.9245) | 38.100 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Uric acid:Week 24, n=5,5,3,1 | 2.570 (10.5697) | -14.008 (11.1139) | -2.893 (5.4966) | 19.050 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 28, n=5,2,3,1: number analyzed (Participants) | 5 | 2 | 3 | 1
  Uric acid:Week 28, n=5,2,3,1 | 2.062 (14.6021) | -6.000 (8.4853) | -6.387 (5.5830) | 33.330 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Uric acid:Week 32, n=4,3,3,1 | 8.103 (17.4601) | 0.243 (27.6106) | -3.767 (9.2418) | 14.290 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 36, n=3,1,3,1: number analyzed (Participants) | 3 | 1 | 3 | 1
  Uric acid:Week 36, n=3,1,3,1 | 0.723 (13.2198) | 42.000 (NA) — Standard deviation could not be calculated for single participant. | -2.957 (6.4150) | 9.520 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 40, n=1,2,2,1: number analyzed (Participants) | 1 | 2 | 2 | 1
  Uric acid:Week 40, n=1,2,2,1 | 3.030 (NA) — Standard deviation could not be calculated for single participant. | 3.970 (36.8120) | -9.580 (1.0748) | 28.570 (NA) — Standard deviation could not be calculated for single participant.
  Uric acid:Week 44, n=1,1,2,0: number analyzed (Participants) | 1 | 1 | 2 | 0
  Uric acid:Week 44, n=1,1,2,0 | -12.120 (NA) — Standard deviation could not be calculated for single participant. | 6.000 (NA) — Standard deviation could not be calculated for single participant. | -1.695 (12.1552) |
  Uric acid:Week 48, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Uric acid:Week 48, n=1,0,1,0 | -6.060 (NA) — Standard deviation could not be calculated for single participant. |  | -20.590 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 52, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Uric acid:Week 52, n=1,0,1,0 | 6.060 (NA) — Standard deviation could not be calculated for single participant. |  | -13.240 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 56, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Uric acid:Week 56, n=1,0,1,0 | -6.060 (NA) — Standard deviation could not be calculated for single participant. |  | -4.410 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 60, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Uric acid:Week 60, n=1,0,1,0 | 9.090 (NA) — Standard deviation could not be calculated for single participant. |  | -1.470 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 64, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Uric acid:Week 64, n=1,0,1,0 | -12.120 (NA) — Standard deviation could not be calculated for single participant. |  | -11.760 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 68, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Uric acid:Week 68, n=1,0,1,0 | -6.060 (NA) — Standard deviation could not be calculated for single participant. |  | -10.290 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Uric acid:Week 72, n=0,0,1,0 |  |  | -11.760 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 76, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Uric acid:Week 76, n=0,0,1,0 |  |  | -20.590 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Uric acid:Week 80, n=0,0,1,0 |  |  | -14.710 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 84, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Uric acid:Week 84, n=0,0,1,0 |  |  | -7.350 (NA) — Standard deviation could not be calculated for single participant. |
  Uric acid:Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Uric acid:Week 88, n=0,0,1,0 |  |  | -17.650 (NA) — Standard deviation could not be calculated for single participant. |

8. Primary Outcome: Percent Change From Baseline in Urine Concentration of Calcium, Creatinine Concentration, Magnesium, Phosphate, Protein During Combination Treatment Period
Description: Urine samples were collected to analyze the urinalysis parameters: Calcium, Creatinine concentration (conc), Magnesium, Phosphate and Protein. Baseline value is the latest GSK2636771 pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Percent change from Baseline was calculated as 100 multiplied by (post-Baseline visit value minus Baseline divided by Baseline).
Time Frame: Baseline (Day 1), Weeks 1, 3, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 48, 56 and 64
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 9 | 7 | 6 | 2
Percent change
  Urine Calcium, Week 1, n=0,0,3,0: number analyzed (Participants) | 0 | 0 | 3 | 0
  Urine Calcium, Week 1, n=0,0,3,0 |  |  | -65.187 (18.5760) |
  Urine Calcium, Week 3, n=8,4,5,1: number analyzed (Participants) | 8 | 4 | 5 | 1
  Urine Calcium, Week 3, n=8,4,5,1 | -17.766 (84.7647) | -46.473 (32.8568) | -54.754 (23.2351) | -95.740 (NA) — Standard deviation could not be calculated for single participant.
  Urine calcium, Week 4, n=6,7,6,2: number analyzed (Participants) | 6 | 7 | 6 | 2
  Urine calcium, Week 4, n=6,7,6,2 | 1.833 (85.3207) | -43.770 (21.3110) | -38.720 (37.1828) | -87.880 (9.6167)
  Urine calcium, Week 8, n=7,6,5,0: number analyzed (Participants) | 7 | 6 | 5 | 0
  Urine calcium, Week 8, n=7,6,5,0 | -22.406 (106.2823) | -39.052 (24.6041) | -38.834 (33.0068) |
  Urine calcium, Week 12, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine calcium, Week 16, n=7,6,3,1: number analyzed (Participants) | 7 | 6 | 3 | 1
  Urine calcium, Week 16, n=7,6,3,1 | -15.649 (92.8636) | -41.387 (16.7494) | -39.437 (47.6551) | -54.050 (NA) — Standard deviation could not be calculated for single participant.
  Urine calcium, Week 20, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine calcium, Week 24, n=5,4,1,1: number analyzed (Participants) | 5 | 4 | 1 | 1
  Urine calcium, Week 24, n=5,4,1,1 | -18.746 (63.7505) | -35.570 (56.9229) | -80.850 (NA) — Standard deviation could not be calculated for single participant. | 32.430 (NA) — Standard deviation could not be calculated for single participant.
  Urine calcium, Week 28, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine calcium, Week 32, n=4,1,1,1: number analyzed (Participants) | 4 | 1 | 1 | 1
  Urine calcium, Week 32, n=4,1,1,1 | -21.723 (80.8076) | -28.700 (NA) — Standard deviation could not be calculated for single participant. | -57.450 (NA) — Standard deviation could not be calculated for single participant. | -70.270 (NA) — Standard deviation could not be calculated for single participant.
  Urine calcium, Week 36, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine calcium, Week 40, n=1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Urine calcium, Week 40, n=1,1,1,1 | 7.690 (NA) — Standard deviation could not be calculated for single participant. | -69.500 (NA) — Standard deviation could not be calculated for single participant. | 3.570 (NA) — Standard deviation could not be calculated for single participant. | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Urine calcium, Week 48, n=1,1,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Urine calcium, Week 48, n=1,1,0,0 | 63.080 (NA) — Standard deviation could not be calculated for single participant. | -69.570 (NA) — Standard deviation could not be calculated for single participant. |  |
  Urine calcium, Week 56, n=1,1,0,0: number analyzed (Participants) | 1 | 1 | 0 | 0
  Urine calcium, Week 56, n=1,1,0,0 | 149.230 (NA) — Standard deviation could not be calculated for single participant. | -42.030 (NA) — Standard deviation could not be calculated for single participant. |  |
  Urine calcium, Week 64, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine calcium, Week 64, n=1,0,0,0 | 13.850 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Creatinine conc, Week 1, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Creatinine conc, Week 3, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Creatinine conc, Week 4, n=3,2,2,0: number analyzed (Participants) | 3 | 2 | 2 | 0
  Urine Creatinine conc, Week 4, n=3,2,2,0 | -4.953 (32.2945) | -2.095 (44.4699) | -28.210 (26.3609) |
  Urine Creatinine conc, Week 8, n=4,2,2,0: number analyzed (Participants) | 4 | 2 | 2 | 0
  Urine Creatinine conc, Week 8, n=4,2,2,0 | -6.328 (17.8300) | -6.815 (21.1071) | -28.420 (14.5947) |
  Urine Creatinine conc, Week 12, n=2,2,2,0: number analyzed (Participants) | 2 | 2 | 2 | 0
  Urine Creatinine conc, Week 12, n=2,2,2,0 | 23.965 (75.8372) | 55.315 (124.3447) | -68.290 (30.3207) |
  Urine Creatinine conc, Week 16, n=1,2,1,0: number analyzed (Participants) | 1 | 2 | 1 | 0
  Urine Creatinine conc, Week 16, n=1,2,1,0 | 87.930 (NA) — Standard deviation could not be calculated for single participant. | -38.040 (15.3725) | -38.920 (NA) — Standard deviation could not be calculated for single participant. |
  Urine Creatinine conc, Week 20, n=3,2,1,0: number analyzed (Participants) | 3 | 2 | 1 | 0
  Urine Creatinine conc, Week 20, n=3,2,1,0 | 34.260 (62.0584) | -56.830 (14.2694) | -56.760 (NA) — Standard deviation could not be calculated for single participant. |
  Urine Creatinine conc, Week 24, n=2,1,0,0: number analyzed (Participants) | 2 | 1 | 0 | 0
  Urine Creatinine conc, Week 24, n=2,1,0,0 | 14.140 (43.4022) | -15.730 (NA) — Standard deviation could not be calculated for single participant. |  |
  Urine Creatinine conc, Week 28, n=3,0,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0
  Urine Creatinine conc, Week 28, n=3,0,0,0 | -39.680 (53.3702) |  |  |
  Urine Creatinine conc, Week 32, n=2,0,0,0: number analyzed (Participants) | 2 | 0 | 0 | 0
  Urine Creatinine conc, Week 32, n=2,0,0,0 | 45.985 (16.6524) |  |  |
  Urine Creatinine conc, Week 36, n=1,0,1,1: number analyzed (Participants) | 1 | 0 | 1 | 1
  Urine Creatinine conc, Week 36, n=1,0,1,1 | 28.450 (NA) — Standard deviation could not be calculated for single participant. |  | 11.350 (NA) — Standard deviation could not be calculated for single participant. | -23.400 (NA) — Standard deviation could not be calculated for single participant.
  Urine Creatinine conc, Week 40, n=0,0,1,1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Urine Creatinine conc, Week 40, n=0,0,1,1 |  |  | -67.570 (NA) — Standard deviation could not be calculated for single participant. | -16.490 (NA) — Standard deviation could not be calculated for single participant.
  Urine Creatinine conc, Week 48, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Creatinine conc, Week 56, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Creatinine conc, Week 64, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Magnesium, Week 1, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Magnesium, Week 3, n=5,3,3,0: number analyzed (Participants) | 5 | 3 | 3 | 0
  Urine Magnesium, Week 3, n=5,3,3,0 | -3.814 (33.8771) | -22.173 (21.2675) | -25.617 (41.4271) |
  Urine Magnesium, Week 4, n=5,4,3,0: number analyzed (Participants) | 5 | 4 | 3 | 0
  Urine Magnesium, Week 4, n=5,4,3,0 | -18.914 (34.9200) | 48.198 (36.5733) | -38.777 (21.3399) |
  Urine Magnesium, Week 8, n=4,4,3,0: number analyzed (Participants) | 4 | 4 | 3 | 0
  Urine Magnesium, Week 8, n=4,4,3,0 | 0.080 (97.5606) | 22.425 (45.1613) | -46.677 (18.8832) |
  Urine Magnesium, Week 12, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Magnesium, Week 16, n=2,3,0,0: number analyzed (Participants) | 2 | 3 | 0 | 0
  Urine Magnesium, Week 16, n=2,3,0,0 | 33.510 (124.1680) | 4.530 (17.5296) |  |
  Urine Magnesium, Week 20, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Magnesium, Week 24, n=3,2,0,0: number analyzed (Participants) | 3 | 2 | 0 | 0
  Urine Magnesium, Week 24, n=3,2,0,0 | -13.997 (66.1097) | 8.425 (50.4804) |  |
  Urine Magnesium, Week 28, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Magnesium, Week 32, n=3,1,0,0: number analyzed (Participants) | 3 | 1 | 0 | 0
  Urine Magnesium, Week 32, n=3,1,0,0 | 4.147 (77.8921) | 82.350 (NA) — Standard deviation could not be calculated for single participant. |  |
  Urine Magnesium, Week 36, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Magnesium, Week 40, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Magnesium, Week 40, n=1,0,0,0 | -77.050 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Magnesium, Week 48, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Magnesium, Week 48, n=1,0,0,0 | 47.540 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Magnesium, Week 56, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Magnesium, Week 56, n=1,0,0,0 | -13.110 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Magnesium, Week 64, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Magnesium, Week 64, n=1,0,0,0 | 19.670 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Phosphate, Week 1, n=0,0,2,0: number analyzed (Participants) | 0 | 0 | 2 | 0
  Urine Phosphate, Week 1, n=0,0,2,0 |  |  | 7.800 (18.9646) |
  Urine Phosphate, Week 3, n=8,4,5,0: number analyzed (Participants) | 8 | 4 | 5 | 0
  Urine Phosphate, Week 3, n=8,4,5,0 | 9.118 (45.4234) | 41.553 (63.8281) | 12.918 (59.9265) |
  Urine Phosphate, Week 4, n=9,6,5,1: number analyzed (Participants) | 9 | 6 | 5 | 1
  Urine Phosphate, Week 4, n=9,6,5,1 | 1.980 (50.5354) | 55.768 (99.4820) | -13.832 (24.3081) | -57.640 (NA) — Standard deviation could not be calculated for single participant.
  Urine Phosphate, Week 8, n=7,7,4,0: number analyzed (Participants) | 7 | 7 | 4 | 0
  Urine Phosphate, Week 8, n=7,7,4,0 | 30.650 (76.2619) | 61.757 (109.4144) | -0.638 (28.7487) |
  Urine Phosphate, Week 12, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Phosphate, Week 16, n=6,5,2,1: number analyzed (Participants) | 6 | 5 | 2 | 1
  Urine Phosphate, Week 16, n=6,5,2,1 | 23.998 (77.8683) | 60.884 (85.7357) | 52.270 (74.6422) | 29.060 (NA) — Standard deviation could not be calculated for single participant.
  Urine Phosphate, Week 20, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Phosphate, Week 24, n=5,3,1,1: number analyzed (Participants) | 5 | 3 | 1 | 1
  Urine Phosphate, Week 24, n=5,3,1,1 | 84.308 (119.7584) | 25.007 (76.8139) | -23.470 (NA) — Standard deviation could not be calculated for single participant. | -0.990 (NA) — Standard deviation could not be calculated for single participant.
  Urine Phosphate, Week 28, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Phosphate, Week 32, n=4,2,1,1: number analyzed (Participants) | 4 | 2 | 1 | 1
  Urine Phosphate, Week 32, n=4,2,1,1 | 48.388 (121.3648) | -22.530 (15.2735) | -2.040 (NA) — Standard deviation could not be calculated for single participant. | -65.020 (NA) — Standard deviation could not be calculated for single participant.
  Urine Phosphate, Week 36, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Phosphate, Week 40, n=1,1,1,1: number analyzed (Participants) | 1 | 1 | 1 | 1
  Urine Phosphate, Week 40, n=1,1,1,1 | 0.000 (NA) — Standard deviation could not be calculated for single participant. | -39.080 (NA) — Standard deviation could not be calculated for single participant. | -3.030 (NA) — Standard deviation could not be calculated for single participant. | -12.320 (NA) — Standard deviation could not be calculated for single participant.
  Urine Phosphate, Week 48, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Phosphate, Week 48, n=1,0,0,0 | 222.220 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Phosphate, Week 56, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Phosphate, Week 56, n=1,0,0,0 | -48.150 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Phosphate, Week 64, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Phosphate, Week 64, n=1,0,0,0 | 37.040 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Protein, Week 1, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Protein, Week 3, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Protein, Week 4, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Urine Protein, Week 4, n=0,1,0,0 |  | -13.790 (NA) — Standard deviation could not be calculated for single participant. |  |
  Urine Protein, Week 8, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Protein, Week 12, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Urine Protein, Week 12, n=0,0,1,0 |  |  | -53.850 (NA) — Standard deviation could not be calculated for single participant. |
  Urine Protein, Week 16, n=0,1,1,0: number analyzed (Participants) | 0 | 1 | 1 | 0
  Urine Protein, Week 16, n=0,1,1,0 |  | -6.900 (NA) — Standard deviation could not be calculated for single participant. | -30.770 (NA) — Standard deviation could not be calculated for single participant. |
  Urine Protein, Week 20, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Urine Protein, Week 20, n=0,0,1,0 |  |  | -53.850 (NA) — Standard deviation could not be calculated for single participant. |
  Urine Protein, Week 24, n=0,1,0,0: number analyzed (Participants) | 0 | 1 | 0 | 0
  Urine Protein, Week 24, n=0,1,0,0 |  | -12.640 (NA) — Standard deviation could not be calculated for single participant. |  |
  Urine Protein, Week 28, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Protein, Week 28, n=1,0,0,0 | -99.430 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Protein, Week 32, n=1,0,0,0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Urine Protein, Week 32, n=1,0,0,0 | -34.780 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Urine Protein, Week 36, n=0,0,1,1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Urine Protein, Week 36, n=0,0,1,1 |  |  | 38.460 (NA) — Standard deviation could not be calculated for single participant. | 33.330 (NA) — Standard deviation could not be calculated for single participant.
  Urine Protein, Week 40, n=0,0,1,1: number analyzed (Participants) | 0 | 0 | 1 | 1
  Urine Protein, Week 40, n=0,0,1,1 |  |  | -53.850 (NA) — Standard deviation could not be calculated for single participant. | 25.000 (NA) — Standard deviation could not be calculated for single participant.
  Urine Protein, Week 48, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Protein, Week 56, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Urine Protein, Week 64, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram (ECG) Findings During Combination Treatment Period
Description: A 12-lead ECG was obtained after the participant had rested at least 5 minutes in a semi-recumbent or supine position at each time point during the study using ECG machine that automatically measured PR, QRS, QT and Corrected QT interval (QT duration corrected for heart rate by Bazett's formula [QTcB] and Fridericia's formula [QTcF]). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Number of participants with abnormal clinical significant ECG findings are presented.
Time Frame: Weeks 4, 8, 16, 24, 32, 40, 48, 56, 64, 72, 80 and 88
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 10 | 9 | 11 | 1
Participants
  Week 4, n=10,8,11,1: number analyzed (Participants) | 10 | 8 | 11 | 1
  Week 4, n=10,8,11,1 | 0 | 0 | 0 | 0
  Week 8, n=8,9,8,0: number analyzed (Participants) | 8 | 9 | 8 | 0
  Week 8, n=8,9,8,0 | 0 | 1 | 1 |
  Week 16, n=8,8,3,1: number analyzed (Participants) | 8 | 8 | 3 | 1
  Week 16, n=8,8,3,1 | 0 | 0 | 0 | 0
  Week 24, n=5,5,3,1: number analyzed (Participants) | 5 | 5 | 3 | 1
  Week 24, n=5,5,3,1 | 0 | 0 | 0 | 0
  Week 32, n=4,3,3,1: number analyzed (Participants) | 4 | 3 | 3 | 1
  Week 32, n=4,3,3,1 | 0 | 0 | 1 | 0
  Week 40, n=1,0,2,1: number analyzed (Participants) | 1 | 0 | 2 | 1
  Week 40, n=1,0,2,1 | 0 |  | 0 | 0
  Week 48, n=1,1,1,0: number analyzed (Participants) | 1 | 1 | 1 | 0
  Week 48, n=1,1,1,0 | 0 | 0 | 0 |
  Week 56, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 56, n=1,0,1,0 | 0 |  | 0 |
  Week 64, n=1,0,1,0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 64, n=1,0,1,0 | 0 |  | 0 |
  Week 72, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Week 72, n=0,0,1,0 |  |  | 0 |
  Week 80, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Week 80, n=0,0,1,0 |  |  | 0 |
  Week 88, n=0,0,1,0: number analyzed (Participants) | 0 | 0 | 1 | 0
  Week 88, n=0,0,1,0 |  |  | 0 |

10. Primary Outcome: Number of Participants With Worst Case Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Results by Maximum Grade Increase Post-Baseline Relative to Baseline During Combination Treatment Period
Description: SBP and DBP were measured after resting for 5 minutes in semi-supine position. SBP and DBP were graded according to Common Toxicity Criteria for Adverse Events (CTCAE) version 4. 'Any grade increase' is defined as an increase in CTCAE grade relative to Baseline grade. For SBP, Grade 0: <120 millimeters of mercury [mmHg]), Grade 1: 120-139 mmHg, Grade 2: 140-159 mmHg, Grade 3:>=160 mmHg. For DBP, Grade 0: <80 mmHg, Grade 1: 80-89 mmHg, Grade 2: 90-99 mmHg, Grade 3: >=100 mmHg. Higher grade indicate worst outcome. Data for worst-case post-Baseline is reported.
Time Frame: Up to maximum 654 days
Population: All Treated Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Participants
  SBP, Any Grade Increase | 8 | 6 | 5 | 1
  SBP, Increase to Grade 2 | 3 | 1 | 3 | 0
  SBP, Increase to Grade 3 | 3 | 2 | 1 | 0
  DBP, Any Grade Increase | 8 | 6 | 5 | 2
  DBP, Increase to Grade 2 | 6 | 4 | 2 | 1
  DBP, Increase to Grade 3 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Worst Case Post-Baseline Results for Heart Rate During Combination Treatment Period
Description: Heart rate was measured after resting for 5 minutes in semi-supine position. The clinical concern range for heart rate was: low: decrease to <60 beats per minute (bpm) and high: increase to >100 bpm. Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'Change to normal or No Change' category. Participants were counted twice if the participant had both values 'decrease to <60 bpm' and 'increase to >100 bpm' during post-Baseline visits. Data for worst case post-Baseline is reported.
Time Frame: Up to maximum 654 days
Population: All Treated Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Participants
  Decrease to <60 | 2 | 2 | 6 | 1
  Change to normal or no change | 8 | 7 | 5 | 1
  Increase to >100 | 1 | 3 | 1 | 1

12. Primary Outcome: Number of Participants With Worst Case Post-Baseline Results for Body Temperature During Combination Treatment Period
Description: Temperature was measured after resting for 5 minutes in semi-supine position. The clinical concern range for body temperature was: low: decrease to <=35 degrees celsius, high: increase to >=38 degrees celsius. Participants were counted in the worst case category that their value changed to (low, within range or no change, or high) unless there was no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became within range, were recorded in the 'Change to normal or No Change' category. Participants were counted twice if the participant had both values 'decreased to <=35 degree celsius' and 'increased to >=38 degrees celsius' during post-Baseline visits. Data for worst-case post-Baseline is presented.
Time Frame: Up to maximum 654 days
Population: All Treated Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 10 | 12 | 2
Participants
  Decrease to <=35 | 0 | 0 | 0 | 0
  Change to normal or no change | 11 | 10 | 10 | 2
  Increase to >=38 | 0 | 0 | 2 | 0

13. Primary Outcome: Non-progressive Disease (Non-PD) Rate at Week 12 According to Prostate Cancer Working Group 2 (PCWG2) Criteria in GSK2636771 200mg/Enzalutamide 160mg - Overall Arm
Description: The 12-week non-PD rate was defined as percentage of participants without progression(non-PD) at Week12 as determined from Prostate-specific antigen(PSA) results, radiographic assessment per Response Evaluation Criteria In Solid Tumors(RECIST)1.1 and bone scan.Disease progression was defined by 1 or more of the following:PSA progression alone; PSA progression according to the PCWG2 criteria with accompanying progression by RECIST1.1 or bone scan for participants with soft tissue Baseline disease; Bone progression on bone scan according to PCWG2 criteria; or Radiographic progression in soft tissue or bone by RECIST1.1 for participants with Baseline disease.Modified All Treated Clinical Activity Population consisted of all participants who received at least 1 dose of GSK2636771 and who were treated at the same dose as dose expansion cohort and have been on study drug for at least 12weeks or have discontinued study treatment due to disease progression, died or withdrawn for any reason.
Time Frame: At Week 12
Population: Modified All Treated Clinical Activity Population. The hypothesis for 12-week non-PD rate was to be tested on a combination of data provided in the dose escalation and dose expansion phase. The 200 mg dose was the only one that had a dose expansion phase. Hence, a combined arm of GSK2636771 200 mg/ Enzalutamide 160 mg has been presented.
Measure: Number; unit: Percentage of participants
Groups:
- GSK2636771 200mg/Enzalutamide 160mg - Overall: Participants received GSK2636771 200 mg with enzalutamide 160 mg either in dose escalation cohort or in dose expansion cohort. This arm contain combined data for dose escalation and dose expansion cohorts of GSK2636771 200 mg/ Enzalutamide 160 mg.
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg - Overall
Number analyzed (Participants) | 22
Percentage of participants | 50

14. Secondary Outcome: Prostate-specific Antigen Decrease From Baseline >=50% (PSA50) Response Rate at 12 Weeks During Combination Treatment Period
Description: PSA50 response rate is defined as percentage of participants with a decrease of >=50% in the PSA concentration from the Baseline PSA value determined at least 12 weeks after start of treatment until last post-treatment follow-up visit or initiation of new anti-cancer therapy and confirmed after 3 or more weeks by an additional PSA evaluation. Confirmed PSA50 is defined as decline of >=50% in PSA concentration from Baseline.
Time Frame: At Week 12
Population: All treated Clinical Activity Population consisted of all participants who received at least one dose of GSK2636771.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Percentage of participants | 9 | 9 | 8 | 50

15. Secondary Outcome: Objective Response Rate (ORR) During Combination Treatment Period
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or a partial response (PR) as the Best Overall Response (BOR), as assessed by the investigator per RECIST Version (v) 1.1 criteria; where CR: Disappearance of all target lesions; PR: at least 30% decrease in the sum of the longest diameter of target lesions with reference to Baseline sum of diameters.
Time Frame: Up to maximum 654 days
Population: All Treated Clinical Activity Population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 2
Percentage of participants
  CR | 0 | 0 | 0 | 0
  PR | 9 | 0 | 0 | 0

16. Secondary Outcome: Time to PSA Progression According to PCWG2 Criteria During Combination Treatment Period
Description: Time to PSA progression is defined as the time from combination study treatment start until the first PSA progression per PCWG2 criteria (confirmed if there has been a PSA decline from Baseline). Time to PSA was analyzed using Kaplan-Meier methods. Median and inter-quartile range (first and third quartile) are presented.
Time Frame: Up to maximum 654 days
Population: All treated Clinical Activity Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 1
Weeks | 19.1 [15.1 to 31.1] | 14.6 [11.3 to 19.1] | 11.4 [11.1 to 19.1] | 11.9 [NA to NA] — As there was a single participant, median value presented is the actual value. Hence, inter quartile range could not be calculated for single participant.

17. Secondary Outcome: Time to Radiological Progression According to PCWG2 Criteria During Combination Treatment Period
Description: Time to radiological progression is defined as the time from combination study treatment start until the first radiological progression by PCWG2 criteria. Time to radiological progession was analyzed using Kaplan-Meier methods. For participants who do not progress, participants were censored at the time of last radiological scan or date of death. Participants who discontinued study with no post-treatment tumor assessment were censored at date of first dose of GSK2636771 drug. Median and inter-quartile range (first and third quartile) are presented.
Time Frame: Up to maximum 654 days
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 1
Weeks | 38.1 [34.3 to 38.1] | 23.1 [11.3 to NA] — <75% of participants experienced the event within the treatment arm and two participants were censored. | 21.9 [14.6 to 43.0] | 38.9 [NA to NA] — As there was a single participant, median value presented is the actual value. Hence, inter quartile range could not be calculated for single participant.

18. Secondary Outcome: Radiological Progression Free Survival (rPFS) Per PCWG2 Criteria During Combination Treatment Period
Description: rPFS is defined as the interval of time (in weeks) between the date of first dose of GSK2636771 and the earlier of the date of disease progression as assessed by the investigator per RECIST version 1.1 criteria and the date of death due to any cause. For participants who do not progress or die, participants were censored at the time of last radiological scan. Participants who discontinued study with no post-treatment tumor assessment were censored at date of first dose of GSK2636771 drug. rPFS was analyzed using Kaplan-Meier methods. Median and inter-quartile range (first and third quartile) are presented.
Time Frame: Up to maximum 654 days
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 11 | 11 | 12 | 1
Weeks | 38.1 [34.3 to 38.1] | 23.1 [11.3 to NA] — <75% of participants experienced the event within the treatment arm and two participants were censored. | 21.9 [14.6 to 43.0] | 38.9 [NA to NA] — As there was a single participant, median value presented is the actual value. Hence, inter quartile range could not be calculated for single participant.

19. Secondary Outcome: Plasma Concentration of GSK2636771 in GSK2636771/Enzalutamide Expansion Cohort in Combination Treatment Period
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2636771.
Time Frame: Week 5: Pre-dose, 1, 2, 3, 5-6, 6-7, 7-8 hours post-dose; Weeks 8 and 12: Pre-dose
Population: Pharmacokinetic Concentration Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Expansion
Number analyzed (Participants) | 7
Nanograms per milliliter
  Week 5: Pre-dose, n=6: number analyzed (Participants) | 6
  Week 5: Pre-dose, n=6 | 4035.000 (2650.9602)
  Week 5: 1 hour, n=6: number analyzed (Participants) | 6
  Week 5: 1 hour, n=6 | 4758.333 (1818.9823)
  Week 5: 2 hours, n=7 | 7124.286 (4328.2362)
  Week 5: 3 hours, n=7 | 9565.714 (4422.4648)
  Week 5: 5-6 hours, n=1: number analyzed (Participants) | 1
  Week 5: 5-6 hours, n=1 | 14600.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 6-7 hours, n=1: number analyzed (Participants) | 1
  Week 5: 6-7 hours, n=1 | 13400.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 7-8 hours, n=1: number analyzed (Participants) | 1
  Week 5: 7-8 hours, n=1 | 14800.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 8: Pre-dose, n=7 | 6291.429 (3742.1492)
  Week 12: Pre-dose, n=6: number analyzed (Participants) | 6
  Week 12: Pre-dose, n=6 | 5328.333 (2756.5879)

20. Secondary Outcome: Plasma Concentration of GSK2636771 in GSK2636771/Enzalutamide Escalation Cohorts in Combination Treatment Period
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK2636771. Pharmacokinetic Concentration Population consisted of all participants in the All Treated Safety Population for whom a blood sample for pharmacokinetics were obtained, analyzed, and was measurable.
Time Frame: Week 5: Pre-dose, 0.5, 1, 2, 3, 4, 6 hours post-dose; Weeks 8 and 12: Pre-dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 8 | 8 | 1
Nanograms per milliliter
  Week 5: Pre-dose, n=8,8,1 | 6720.000 (3376.1136) | 5142.500 (1613.1402) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 0.5 hours, n=8,6,1: number analyzed (Participants) | 8 | 6 | 1
  Week 5: 0.5 hours, n=8,6,1 | 8059.250 (4085.9045) | 5008.333 (1170.4771) | 292.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 1 hours, n=7,7,1: number analyzed (Participants) | 7 | 7 | 1
  Week 5: 1 hours, n=7,7,1 | 8620.714 (4561.6832) | 5794.286 (994.8175) | 433.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 2 hours, n=8,8,1 | 8811.875 (4424.590) | 8408.750 (1764.7374) | 3510.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 3 hours, n=8, 8,1 | 9776.875 (4869.5519) | 10510.000 (3375.0725) | 6690.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 4 hours, n=7,8,1: number analyzed (Participants) | 7 | 8 | 1
  Week 5: 4 hours, n=7,8,1 | 8921.429 (4857.7959) | 11250.000 (3639.5172) | 9060.000 (NA) — Standard deviation could not be calculated for single participant.
  Week 5: 6 hours, n=6,8,0: number analyzed (Participants) | 6 | 8 | 0
  Week 5: 6 hours, n=6,8,0 | 7264.833 (4319.3051) | 10073.750 (3000.0664) |
  Week 8: Pre-dose, n=7,6,0: number analyzed (Participants) | 7 | 6 | 0
  Week 8: Pre-dose, n=7,6,0 | 9354.286 (3676.1477) | 7333.333 (4236.7802) |
  Week 12: Pre-dose, n=6,5,0: number analyzed (Participants) | 6 | 5 | 0
  Week 12: Pre-dose, n=6,5,0 | 7938.333 (3801.3756) | 8036.000 (3025.3479) |

21. Secondary Outcome: Plasma Concentration of Enzalutamide in GSK2636771/Enzalutamide Escalation Cohorts in Combination Treatment Period
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of enzalutamide.
Time Frame: Week 5: Pre-dose, 0.5, 1, 2, 3, 4, 6 hours post-dose; Weeks 8 and 12: Pre-dose
Population: Pharmacokinetic Concentration Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles). Blood samples were not collected for analysis of Enzalutamide for GSK2636771 400mg/Enzalutamide 160mg Escalation arm.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 9 | 7 | 0
Micrograms per milliliter
  Week 5: Pre-dose, n=9,7,0 | 12.131 (3.0795) | 12.134 (3.2382) |
  Week 5: 0.5 hours, n=9,6,0: number analyzed (Participants) | 9 | 6 | 0
  Week 5: 0.5 hours, n=9,6,0 | 14.178 (2.4929) | 13.545 (3.9395) |
  Week 5: 1 hours, n=7,7,0: number analyzed (Participants) | 7 | 7 | 0
  Week 5: 1 hours, n=7,7,0 | 14.771 (2.8224) | 14.829 (2.7980) |
  Week 5: 2 hours, n=9,7,0 | 13.611 (3.5674) | 14.200 (2.7761) |
  Week 5: 3 hours, n=8,7,0: number analyzed (Participants) | 8 | 7 | 0
  Week 5: 3 hours, n=8,7,0 | 14.600 (3.4748) | 12.586 (2.8416) |
  Week 5: 4 hours, n=9,7,0 | 12.536 (3.3727) | 12.466 (3.4905) |
  Week 5: 6 hours, n=7,7,0: number analyzed (Participants) | 7 | 7 | 0
  Week 5: 6 hours, n=7,7,0 | 11.741 (3.0012) | 12.150 (3.6842) |
  Week 8: Pre-dose, n=5,5,0: number analyzed (Participants) | 5 | 5 | 0
  Week 8: Pre-dose, n=5,5,0 | 13.140 (2.7337) | 12.240 (2.1126) |
  Week 12: Pre-dose, n=4,4,0: number analyzed (Participants) | 4 | 4 | 0
  Week 12: Pre-dose, n=4,4,0 | 12.333 (3.8684) | 12.750 (1.6176) |

22. Secondary Outcome: Plasma Concentration of Enzalutamide in GSK2636771/Enzalutamide Expansion Cohort in Combination Treatment Period
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of enzalutamide.
Time Frame: Week 5: Pre-dose, 1, 2, 3, 5-6, 6-7, 7-8 hours post-dose; Weeks 8 and 12: Pre-dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Expansion
Number analyzed (Participants) | 8
Micrograms per milliliter
  Week 5: Pre-dose, n=6: number analyzed (Participants) | 6
  Week 5: Pre-dose, n=6 | 11.735 (2.3463)
  Week 5: 1 hour, n=7: number analyzed (Participants) | 7
  Week 5: 1 hour, n=7 | 14.793 (3.8293)
  Week 5: 2 hours, n=7: number analyzed (Participants) | 7
  Week 5: 2 hours, n=7 | 13.274 (2.9788)
  Week 5: 3 hours, n=7: number analyzed (Participants) | 7
  Week 5: 3 hours, n=7 | 12.886 (4.1615)
  Week 5: 5-6 hours, n=2: number analyzed (Participants) | 2
  Week 5: 5-6 hours, n=2 | 13.800 (0.7071)
  Week 5: 6-7 hours, n=2: number analyzed (Participants) | 2
  Week 5: 6-7 hours, n=2 | 13.300 (1.4142)
  Week 5: 7-8 hours, n=2: number analyzed (Participants) | 2
  Week 5: 7-8 hours, n=2 | 12.750 (0.3536)
  Week 8: Pre-dose, n=8 | 11.335 (2.5525)
  Week 12: Pre-dose, n=6: number analyzed (Participants) | 6
  Week 12: Pre-dose, n=6 | 11.520 (3.1956)

23. Secondary Outcome: Plasma Concentration of N-desmethyl Enzalutamide in GSK2636771/Enzalutamide Escalation Cohorts in Combination Treatment Period
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of N-desmethyl enzalutamide.
Time Frame: Week 5: Pre-dose, 0.5, 1, 2, 3, 4, 6 hours post-dose; Weeks 8 and 12: Pre-dose
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
Number analyzed (Participants) | 9 | 7 | 0
Micrograms per milliliter
  Week 5: Pre-dose, n=9,7,0 | 13.057 (3.5612) | 12.583 (4.4768) |
  Week 5: 0.5 hours, n=9,6,0: number analyzed (Participants) | 9 | 6 | 0
  Week 5: 0.5 hours, n=9,6,0 | 13.257 (3.0229) | 12.208 (4.9689) |
  Week 5: 1 hours, n=7,7,0: number analyzed (Participants) | 7 | 7 | 0
  Week 5: 1 hours, n=7,7,0 | 12.736 (2.6587) | 11.350 (4.4129) |
  Week 5: 2 hours, n=9,7,0 | 11.710 (2.7646) | 11.449 (3.9828) |
  Week 5: 3 hours, n=8,7,0: number analyzed (Participants) | 8 | 7 | 0
  Week 5: 3 hours, n=8,7,0 | 13.189 (2.5728) | 11.136 (4.4445) |
  Week 5: 4 hours, n=9,7,0 | 11.426 (2.1615) | 10.703 (3.5853) |
  Week 5: 6 hours, n=7,7,0: number analyzed (Participants) | 7 | 7 | 0
  Week 5: 6 hours, n=7,7,0 | 11.256 (2.6641) | 10.416 (1.7444) |
  Week 8: Pre-dose, n=5,5,0: number analyzed (Participants) | 5 | 5 | 0
  Week 8: Pre-dose, n=5,5,0 | 14.200 (1.7450) | 13.348 (4.4348) |
  Week 12: Pre-dose, n=4,4,0: number analyzed (Participants) | 4 | 4 | 0
  Week 12: Pre-dose, n=4,4,0 | 13.665 (5.3833) | 11.958 (2.4890) |

24. Secondary Outcome: Plasma Concentration of N-desmethyl Enzalutamide in GSK2636771/Enzalutamide Expansion Cohort in Combination Treatment Period
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of N-desmethyl enzalutamide.
Time Frame: Week 5: Pre-dose, 1, 2, 3, 5-6, 6-7, 7-8 hours post-dose; Weeks 8 and 12: Pre-dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | GSK2636771 200mg/Enzalutamide 160mg Expansion
Number analyzed (Participants) | 8
Micrograms per milliliter
  Week 5: Pre-dose, n=6: number analyzed (Participants) | 6
  Week 5: Pre-dose, n=6 | 11.623 (3.5552)
  Week 5: 1 hour, n=7: number analyzed (Participants) | 7
  Week 5: 1 hour, n=7 | 12.476 (3.6642)
  Week 5: 2 hours, n=7: number analyzed (Participants) | 7
  Week 5: 2 hours, n=7 | 12.069 (3.9492)
  Week 5: 3 hours, n=7: number analyzed (Participants) | 7
  Week 5: 3 hours, n=7 | 11.861 (4.1782)
  Week 5: 5-6 hours, n=2: number analyzed (Participants) | 2
  Week 5: 5-6 hours, n=2 | 11.850 (0.3536)
  Week 5: 6-7 hours, n=2: number analyzed (Participants) | 2
  Week 5: 6-7 hours, n=2 | 11.135 (2.7789)
  Week 5: 7-8 hours, n=2: number analyzed (Participants) | 2
  Week 5: 7-8 hours, n=2 | 11.050 (2.8991)
  Week 8: Pre-dose, n=8 | 14.450 (4.7827)
  Week 12: Pre-dose, n=6: number analyzed (Participants) | 6
  Week 12: Pre-dose, n=6 | 15.690 (7.4271)

ADVERSE EVENTS:
Time Frame: Up to Week 2 for run-in period and up to maximum of 675 days for combination treatment period
Description: All Treated Safety Population consisted of all participants who received at least one dose of GSK2636771 or Enzalutamide.
Arm/Group | Enzalutamide Only (run-in Period) | GSK2636771 200mg/Enzalutamide 160mg Escalation | GSK2636771 200mg/Enzalutamide 160mg Expansion | GSK2636771 300mg/Enzalutamide 160mg Escalation | GSK2636771 400mg/Enzalutamide 160mg Escalation
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/11 | 0/11 | 0/12 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/37 | 2/11 | 2/11 | 2/12 | 0/2
Other Adverse Events (participants affected / at risk) | 11/37 | 11/11 | 11/11 | 12/12 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide Only (run-in Period) (N=37) | GSK2636771 200mg/Enzalutamide 160mg Escalation (N=11) | GSK2636771 200mg/Enzalutamide 160mg Expansion (N=11) | GSK2636771 300mg/Enzalutamide 160mg Escalation (N=12) | GSK2636771 400mg/Enzalutamide 160mg Escalation (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide Only (run-in Period) (N=37) | GSK2636771 200mg/Enzalutamide 160mg Escalation (N=11) | GSK2636771 200mg/Enzalutamide 160mg Expansion (N=11) | GSK2636771 300mg/Enzalutamide 160mg Escalation (N=12) | GSK2636771 400mg/Enzalutamide 160mg Escalation (N=2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (10) | 8 (19) | 7 (7) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 4 (5) | 5 (5) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 4 (5) | 4 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 1 (1) | 5 (5) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 5 (7) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (2) | 3 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood parathyroid hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroxine decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT02215096/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT02215096/SAP_001.pdf